'-1--'--1 A --1 --'- DI

| Statistical and Epidemiological Analysis Plan | |
|---|---|
| BI Study No.: | 1245.97 |
| Title: | Post-authorisation safety study to assess the risk of urinary tract malignancies in relation to empagliflozin exposure in patients with type 2 diabetes: a multi-database European study |
| Responsible statistician: | and |
| Responsible project epidemiologist: | (principal investigator). |
| Date of statistical and epidemiological analysis plan: | 26-JUL-2022 |
| Version: | 6.0 |
| | Proprietary confidential information im International GmbH or one or more of its affiliated companies. All rights reserved. or in part - be passed on, reproduced, published or otherwise used without prior written permission. |

## **TABLE OF CONTENTS**

| <b>TABL</b> | <b>E OF CONTENTS</b> | 2 |
|-------------|-----------------------------------------------|----|
| | OF ABBREVIATIONS | |
| LIST ( | OF TABLES | 7 |
| 1. | INTRODUCTION | 10 |
| 2. | RESEARCH QUESTION AND OBJECTIVES | 11 |
| 2.1. | RESEARCH QUESTION | 11 |
| 2.2. | OBJECTIVES | |
| 3. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY. | |
| 4. | RESEARCH METHODS | 17 |
| 4.1. | STUDY DESIGN | |
| 4.2. | SETTING | 18 |
| 4.2.1. | STUDY POPULATIONS | 18 |
| 4.2.2. | STUDY PERIOD | |
| 4.2.3. | BASELINE AND LOOK-BACK PERIOD | 18 |
| 4.2.4. | INCLUSION AND EXCLUSION CRITERIA | 20 |
| <b>5.</b> | VARIABLES | 24 |
| 5.1. | EXPOSURES | 24 |
| 5.1.1. | STUDY MEDICATIONS | 24 |
| 5.1.2. | INDEX DATE | 24 |
| 5.1.3. | EXPOSURE TIME | 24 |
| 5.1.4. | DAYS' SUPPLY AND DURATION OF EXPOSURE | 27 |
| 5.1.5. | DOSE 29 | |
| 5.1.6. | DEFINITION OF CONTINUOUS TREATMENT AND | |
| | DISCONTINUATION | 29 |
| 5.1.7. | PRIMARY EXPOSURE DEFINITION | 29 |
| 5.1.8. | SECONDARY EXPOSURE DEFINTIONS | 30 |
| <b>5.2.</b> | OUTCOMES | 31 |
| 5.2.1. | PRIMARY OUTCOMES | 31 |
| 5.3. | COVARIATES | 35 |
| 5.3.1. | DEMOGRAPHICS AND OTHER BASELINE VARIABLES | 35 |
| 5.3.2. | CONCOMITANT DISEASES | 38 |
| 5.3.3. | CONCOMITANT MEDICATIONS | |
| 6. | PLANNED ANALYSIS | 48 |
| 6.1. | SUMMARY OF STUDY POPULATION IDENTIFICATION | |
| <b>6.2.</b> | POPULATION DESCRIPTION BEFORE MATCHING | 49 |
| 6.3. | METHODS ADDRESSING BIAS | 49 |
| 64 | | |

| <b>6.5.</b> | IMPLEMENTATION OF THE PROPENSITY SCORE |
|-------------|------------------------------------------------|
| | MATCHING50 |
| 6.5.1. | ESTIMATION OF THE PROPENSITY SCORE50 |
| 6.5.2. | MATCHING METHOD51 |
| 6.6. | ASSESSING THE QUALITY OF THE MATCHING52 |
| 6.6.1. | PROPENSITY SCORE DISTRIBUTION BEFORE AND AFTER |
| | MATCHING AND COMMON SUPPORT REGION52 |
| 6.6.2. | ASSESSMENT OF COVARIATE BALANCE BEFORE AND |
| | <b>AFTER MATCHING52</b> |
| <b>6.7.</b> | AS-TREATED ANALYSIS53 |
| 6.7.1. | DESCRIPTIVE ANALYSIS53 |
| 6.7.2. | COMPARATIVE ANALYSIS55 |
| 6.7.3. | META-ANALYSES56 |
| 6.7.3. | I. META-ANALYSIS OF DESCRIPTIVE ANALYSES56 |
| 6.7.3.2 | 2. META-ANALYSIS OF COMPARATIVE ANALYSIS57 |
| 6.10. | LIST OF PLANNED ANALYSIS68 |
| 7. | DATA MANAGEMENT78 |
| 8. | STATISTICAL SOFTWARE78 |
| 9. | |
| | QUALITY CONTROL78 |
| | REFERENCES80 |
| | EX I DIAGNOSIS AND OPERATION CODES81 |
| | EX II ATC CODES USED TO DEFINE TREATMENTS83 |
| ANNI | EX III TABLES AND FIGURES TEMPLATES87 |
| ANNI | EX IV LIST OF DRUG DOSAGES FOR EMPAGLIFLOZIN, |
| | DPP-4 INHIBITORS AND METFORMIN185 |

## LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| AT | As-treated analysis |
| ATC | Anatomical Therapeutic Chemical Classification System |
| AvoHILMO | Register of Primary Health Care Visits (Finland) |
| BI | Boehringer Ingelheim International GmbH |
| BMI | Body mass index |
| CI | Confidence interval |
| CLR | Conditional logistic regression |
| COPD | Chronic obstructive pulmonary disease |
| CPRD-GOLD | Clinical Practice Research Datalink, General practitioner OnLine Data (United Kingdom) |
| CPRD Aurum | Clinical Practice Research Datalink, Aurum (United Kingdom) |
| DPP-4 | Dipeptidyl peptidase-4 |
| eGFR | Estimated glomerular filtration rate |
| EMA | European Medicines Agency |
| ENCePP | European Network of Centres for Pharmacoepidemiology and Pharmacovigilance |
| EU | European Union |
| FCR | Finnish Cancer Registry |
| FDA | Food and Drug Administration |
| FPR | Finnish Prescription Register |
| GLP-1 | Glucagon-like peptide-1 |
| GP | General practitioner |
| GPP | Good Pharmacoepidemiology Practices |
| GPV | Good Pharmacovigilance Practices |
| HbA1c | Glycated hemoglobin A1c |
| HES | Hospital Episode Statistics (United Kingdom) |
| HF | Heart failure |
| HILMO | Care Register for Health Care (secondary care; Finland) |
| HR | Hazard ratio |
| ICD-10 | International classification of diseases |

# SEAP for non-interventional study BI Study No: 1245.97

| Term | Definition / description |
|---|---|
| IPTW | Inverse-probability of treatment weights |
| IR | Incidence rate |
| ITT | Intention-to-treat analysis |
| LISA | Longitudinal integration database for health insurance and labour market studies |
| MDRD | Modification of Diet in Renal Disease study |
| MI | Myocardial infarction |
| MSM | Marginal structural model |
| NCC | Nested case-control |
| NDR | National diabetes register (Sweden) |
| NHS | National Health Service |
| NICE | National Institute for Health and Care Excellence |
| NPR | National patient register (Sweden) |
| NSAID | Non-steroidal anti-inflammatory drugs |
| ONS | Office for National Statistics |
| PASS | Post-safety study |
| PH | Proportional hazards |
| PID | Personal identification number |
| PRAC | Pharmacovigilance Risk Assessment Committee |
| PS | Propensity score |
| PSUR | Periodic Safety Update Report |
| PY | Person-years |
| RMP | Risk management plan |
| RR | Relative risk |
| SCR | Swedish cancer registry |
| SEAP | Statistical/Epidemiological Analysis Plan |
| SF | Statistics Finland |
| SGLT-2 | Sodium glucose co-transporter-2 |
| SID | Study identification number |
| SII | Social Insurance Institution (SII) |
| SIR | Standardized incidence ratio |

# SEAP for non-interventional study BI Study No: 1245.97

| Term | Definition / description |
|------|-----------------------------------------------------|
| SPDR | Swedish prescribed drug register |
| T2DM | Type 2 diabetes mellitus |
| THIN | The Health Improvement Network database |
| THL | National Institute for Health and Welfare (Finland) |
| UK | United Kingdom |
| US | United States |
| UT | Urinary tract |
| UTI | Urinary tract infection |

# LIST OF TABLES

| Table 1 Data sources with look-back periods and total data collection periods | 19 |
|---|---|
| Table 2 Inclusion criteria. | 20 |
| Table 3 Exclusion criteria. | 22 |
| Table 4 Censoring events | 26 |
| Table 5 As-treated exposure definition. | 30 |
| Table 6 Exposure definitions based on dosage or duration | 30 |
| Table 7 Intention-to-treat exposure definition. | 31 |
| Table 8 Main outcomes | 32 |
| Table 11 Demographics and other baseline variables | 35 |
| Table 12 Diabetic complications variables. | 38 |
| Table 13 Other non-diabetic concomitant disease variables | 41 |
| Table 14 Other diabetic medication exposure definitions. | 45 |
| Table 15 Other non-diabetic concomitant medication use variables. | 47 |
| Table 16 List of planned analyses. | 68 |
| Table 17 Patients baseline characteristics in each of the study groups and in the total stupopulation in [Study country]. | |
| Table 18 Covariate balance assessment [before/after] matching comparing empagliflozing group to DPP-4 inhibitors group – [Study country] | |
| Table 19 Propensity score distribution before and after propensity score matching of empagliflozin users and DPP-4 inhibitors users by decile in [country] | 119 |
| Table 20 Number of patients with incidence of cancer within 12 months after index date | 120 |
| Table 21 TNM staging of [Study outcome] at diagnosis during follow-up after exclusion cancers occurring within 6 months after index date. | |
| Table 22 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country/pooled] matched cohort(s). The number of patients in strata and the total number of person years are also presented | n each |
| Table 23 Crude hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table show hazard ratios (HRs) using the crude model with the corresponding 95% CI and p-va As treated | alue– |
| Table 24 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Coxproportional hazards model in the [Study country] matched cohort. The table shows | |

| Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|
| hazard ratios (HRs) using the base model with the corresponding 95% CI and p-value— As treated exposure definition |
| Table 25 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—As treated exposure definition. [Stratifying variable if any] |
| Table 26 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—Cumulative dose of empagliflozin exposure definition |
| Table 27 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—daily dose of empagliflozin exposure definition |
| Table 28 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—Cumulative exposure duration to empagliflozin |
| Table 29 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented |
| Table 30 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented |
| Table 31 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented |
| Table 32 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented |
| Table 36. Number of yearly albuminaria tests stratified by exposure group - [Study country] |

| Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|
| Table 37 Patients baseline characteristics in each of the study groups in the UK, stratified by CPRD database |
| Table 38 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the UK-CPRD population stratified by CPRD databases (GOLD and Aurum) . The number of patients in each strata and the total number of person years are also presented |
| Table 39 Crude hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort, stratified by databases. The table shows the hazard ratios (HRs) using the crude model with the corresponding 95% CI and p-value—As treated |
| Table 40 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort, stratified by databases. The table shows the hazard ratios (HRs) using the base model with the corresponding 95% CI and p-value—As treated |
| Table 41 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort, stratified by databases. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—As treated |
| Table 42 Crude hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort after adding CPRD database as a stratification variable. The table shows the hazard ratios (HRs) using the crude model with the corresponding 95% CI and p-value—As treated |
| Table 43 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort after adding CPRD database as a stratification variable. The table shows the hazard ratios (HRs) using the base model with the corresponding 95% CI and p-value—As treated exposure definition |
| Table 44 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort after adding CPRD database as a stratification variable. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—As treated exposure definition. |
| Table 45. Incidence rate of urinary tract cancer in the source population for study years 2015-2020 |

#### 1. INTRODUCTION

This statistical analysis plan refers to the final version of the pharmacoepidemiological study protocol entitled "Post-authorisation safety study to assess the risk of urinary tract malignancies in relation to empagliflozin exposure in patients with type 2 diabetes: a multi-database European study", version 6.0 dated February 10<sup>th</sup>, 2022 unless otherwise stated.

This is an observational, comparative cohort safety study based on European healthcare databases and includes databases from the UK, Sweden and Finland.

The study will use a new user design to compare new users of empagliflozin to new users of DPP-4 inhibitors in order to assess the risk of urinary tract malignancies.

Individuals with similar treatment and clinical history will be matched by deriving propensity scores conditional on factors potentially affecting the treatment and outcome.

In the primary analysis, propensity-score (PS) matched cohorts will be derived from the study base by matching patients who initiate empagliflozin with patients who initiate DPP-4 inhibitors at index date with a variable matching ratio of up to 1:3 (1:1 matching in a sensitivity analysis) using greedy matching methods.

In addition, patients using metformin in free or fixed dose combination with empagliflozin or with a DPP-4 inhibitor will be identified and the primary analysis will be repeated within this subset of patients.

## 2. RESEARCH QUESTION AND OBJECTIVES

## 2.1. RESEARCH QUESTION

The aim of the study is to assess the risk of urinary tract malignancies in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor.

#### 2.2. OBJECTIVES

### **Primary objectives**

- i. To estimate the adjusted hazard ratio and incidence rates of all urinary tract cancers (bladder, renal and other urinary tract cancers) in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor.
- ii. To estimate the adjusted hazard ratios and incidence rates of bladder cancer in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor.
- iii. To estimate the adjusted hazard ratios and incidence rates of renal cancer in patients initiating empagliflozin compared to patients initiating a DPP-4 inhibitor.

#### **Secondary objectives**

- i. To estimate the adjusted hazard ratio and incidence rates of each primary outcome (all urinary tract cancers, bladder cancer, renal cancer) with respect to:
  - a. Increasing cumulative dosage to empagliflozin.
  - b. Dosage of empagliflozin prescribed per use (10mg vs. 25mg).
  - c. Time since first prescribed/dispensed dose of empagliflozin.



## 3. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

| No. | Date | Section of the SEAP | Amendment or update | Reason |
|---|---|---|---|---|
| 1 | 13-October-<br>2017 | Interim<br>reports | Use of patient level data for the 2 <sup>nd</sup> and 3 <sup>rd</sup> interim reports instead of aggregated data. | PRAC assessment comments on the the 1 <sup>st</sup> interim report. |
| 2 | 29-NOV-2019 | Multiple | Inclusion of new study country, Finland. | To increase of the size of the patient population |
| 3 | 29-NOV-2019 | Multiple | Using DPP-4 inhibitors as the primary comparison group and other SGLT-2 inhibitors as the secondary comparison group. | Comparison with other SGLT-2 inhibitors is expected to be underpowered due to the low uptake of SGLT-2 inhibitors other than empagliflozin. The number of patients initiating SGLT-2 inhibitors other than empagliflozin and verifying the inclusion and exclusion criteria in both study countries between August 1st, 2014 and November 30th, 2018 was 10,528 subjects. In contrast, the corresponding number of eligible patients initiating DPP-4 inhibitors was 3.8 times higher than the number of empagliflozin patients with 67,511 subjects. |
| 4 | 29-NOV-2019 | Multiple | Extending the study period until 31 December 2020. | Increasing the study sample size and accounting for the long latency period related to risk of malignancies |
| 5 | 29-NOV-2019 | Multiple | Investigation of patients counts in CPRD Aurum. | Based on the results of the PRAC feasibility evaluation, the number of persons available in CPRD-Aurum will be monitored. |

| 6 | 13-APR-2022 | Multiple | Removal of SGLT-2 inhibitors as a secondary comparator group | Low uptake of SGLT-2 inhibitors other than empagliflozin was observed in the 5 <sup>th</sup> interim report. The number of patients initiating SGLT-2 inhibitors other than empagliflozin and verifying the inclusion and exclusion criteria during the study period was lower than the number of similar patients initiating empagliflozin in Sweden and Finland. It would therefore not be possible to carry out even 1:1 matching for empaglifozin users. |
|---|---|---|---|---|
| 7 | 13-APR-2022 | 6.5 | Change of the PS matching ratio to up to 1:3 matheing in the main analysis and to 1:1 matching in a sensitivity analysis. | Up to 1:3 matching will allow an optimal use of available DPP-4 initiators. Using as many matches as possible in ech country will increase study precision and statistical power. |
| 8 | 13-APR-2022 | 6.7.2 | The description of the Crude, base and fullly adjusted models was aligned with the protocol. Additional criteria for selecting covariates for adjustement were introduced. | The incidence rates observed in the 5 <sup>th</sup> interim report suggest there will be few events for outcomes such as renal cancer. With few events, it will not be possible to build a model including all selected confounders. The chosen method limits the covariates of the model to confounders which are not balanced in the matched sample. |

| 9 | 13-APR-2022 | Multiple | Pooled analysis of individual level data are replaced with aggregate level data meta-analyses. Pooled IRs will be estimated by pooling aggregate level data. Pooled HRs will be estimated using meta-analysis methods. | Individual level data from Finland and Sweden cannot be pooled together due to new regulations in the storage and use of individual level data in Sweden and Finland. |
|---|---|---|---|---|
| 10 | 13-APR-2022 | Multiple | Covariate selection criteria were added to mitigate the effect of missing data as well as potential Cox model convergence failures due to small number of events. | Observed incidence rates in interim report 5 suggests that there will be very few events observed for some outcomes such as renal cancer. In addition, stratified analyses that were to be carried out on pooled individual data will now be carried out at the single country level. It is therefore necessary to plan for possible convergence failure for some Cox proportional hazards models. |

| | | | Specified algorihhms for inclusion and exclusion criteria | |
|---|---|---|---|---|
| | | | Redefined the AT and ITT exposure definitions as two time-fixed variables | |
| | | | Adjusted the definitions of time at risk, latency period and treatment discontinuation. | Modifications made to |
| 12 | 13-APR-2022 | Multiple | Specified algorithms for drug exposure definitions. | clarify the expected analyses for programmers. |
| | | | Removed stratification of metformin use from stratified analyses. (Analyses in study groups have covered subgroups by metformin use) | |
| | | | Changed some covariates from time-dependent to time-fixed | |
| 13 | 13-APR-2022 | Multiple | Sections and tables shells relating to analyses only relevant for interim reports were removed. | This SAP will be used for the final analysis only. |
| 14 | 13-APR-2022 | 6.8.3 | Added sensitivity analysis for grace period | The sensitivity analysis will assess the effect of lengthening the grace period to 90 days. |
| | | | PS variable "database" added for UK CPRD | The CPRD Aurum database |
| 15 | 26 JUL 2022 | Multiple | Additional sensitivity<br>analyses added for UK<br>CPRD | was added to the study upon PRAC request. |

# Boehringer Ingelheim

SEAP for non-interventional study BI Study No: 1245.97 

| 16 | 26 JUL 2022 | Multiple | Extending the study period until 31 December 2021 for UK CPRD-GOLD and Aurum. | Increasing the study sample size and accounting for the long latency period related to risk of malignancies |
|---|---|---|---|---|
|---|---|---|---|---|

#### 4. RESEARCH METHODS

#### 4.1. STUDY DESIGN

This is a non-interventional, comparative, cohort safety study based on European healthcare databases and includes databases from the UK, Sweden and Finland. The databases for this study are constructed from linked prescription, hospital, general practitioner, cancer and death registration records.

The study will use an "incident users" design and compare new users of empagliflozin to new users of DPP-4 inhibitors. The index date will be defined as the date on which each identified new user receives the index prescription for empagliflozin, or a DPP-4 inhibitor.

To minimize channelling bias, individuals will be matched with similar treatment and clinical history at index date by deriving propensity scores (PS) conditional on factors affecting the treatment and outcome [1], [2]. Propensity-score-matched cohorts will be derived from the study base by matching patients who initiate empagliflozin with patients who initiate DPP-4 inhibitors at index date with the highest possible matching ratio (1:1, 1:2, or 1:3 using Greedy matching methods).

Depending on sample size, combination exposures with metformin will be accounted for through separate PS, stratification, or adjustment. Additional analyses will explore the presence of detection/diagnostic bias as screening for urinary tract signs or symptoms may be more frequently among empagliflozin users. The potential for diagnostic bias will be evaluated and addressed through consideration of the frequency of urine dipstick testing (as captured through albuminuria tests) and stage of cancer at the time of diagnosis (as more early-stage cancers in one group would be suggestive of diagnostic bias).

The primary, secondary, and further analyses utilize a cohort design which will allow direct estimation of the IRs and aHRs of multiple outcomes of interest among new users of empagliflozin compared with new users of a DPP-4 inhibitor. The covariate information will be assessed during the time preceding treatment initiation (varying length look-back (preindex) period) and during follow-up and will include all historical information available for each patient up until occurrence of outcome or censoring. Follow-up will start 6 months after the index date (12 months in sensitivity analyses) to account for an empirical induction/promotion period.

In the context of data sources such as the CPRD and the Swedish and Finnish national registers, the use of a cohort design has more advantages than limitations compared with the use of a nested case-control (NCC) design—see the appendix discussion in Schneeweiss (2010) [1] and Patorno et al. (2014) [2]. Thus, an observational cohort is constructed to study the risk of urinary tract malignancies among the two treatment groups. Several sensitivity analyses will be conducted including analyses using a NCC design (given the rarity of the outcomes) and analyses using marginal structural models (MSM) to control for time-varying confounderstowards switching or discontinuation of primary exposure.

The country-level datasets will be analysed separately. Country-level effect size estimates (IRs, aHRs, etc) will be pooled using suitable meta-analysis methods to compute overall estimates.

#### **4.2. SETTING**

#### 4.2.1. STUDY POPULATIONS

The broad study population, in each of the study countries (see data sources in Table 1), will include individuals who have purchased at least one prescription of empagliflozin or of a DPP-4 inhibitor between 1st August, 2014 and 31st December, 2020 (31st December 2021 for UK-CPRD).

The Swedish prescribed drug register (SPDR) and the Finnish prescription register (FPR) will be used to identify the source population in Sweden and Finland. The CPRD-GOLD and CPRD Aurum data will be used to identify the source population in the UK [3]. Patients belonging to a practice having moved from GOLD to Aurum will be present in data extracted from both CPRD-GOLD and Aurum. These patients will be identified using a migrating practices file and their data will be removed from the extracted CPRD-GOLD data. Data from GOLD and Aurum will be combined and treated as a single data source.

ATC codes for empagliflozin and DPP-4 inhibitors are provided in Annex II.

#### 4.2.2. STUDY PERIOD

The study will include individuals who have purchased at least one prescription of empagliflozin or of DPP-4 inhibitors from 1st August 2014 through 31st December 2020 (31st December 2021 for UK-CPRD data). The start of the study period corresponds to the time of drug licensing (second half of 2014 in all three countries) and subsequent introduction into clinical practice. The maximum follow-up time for an individual will be six years.

## 4.2.3. BASELINE AND LOOK-BACK PERIOD

To characterize the empagliflozin and DPP-4 inhibitor cohorts at the time of study drug initiation, all information available during the look-back (pre-index) time period will be collected.

The look-back time period is defined as the time period ending on the day before the index date (Table 1). Since all cohort members are required by inclusion criteria to have at least 1 year of data before the index date (baseline period), the look-back period will include at least 365 days during which covariates can be evaluated. For some study participants, data on covariates might be available beyond 1 year prior to the index date; in these cases, all available information will be considered for covariate classification related to diabetes, diabetes medications, and concomitant chronic conditions. For concomitant medications for diseases other than diabetes, the look-back time period will be limited to 180 days prior to the index date.

Table 1 Data sources with look-back periods and total data collection periods.

| Data source | Data holder | Look-back<br>period | Total data collection period |
|---|---|---|---|
| United Kingdom (UK) | • | | • |
| Clinical Practice Research<br>Datalink, General practitioner<br>OnLine Data (CPRD-GOLD) | Clinical Practice Research<br>Datalink (CPRD) | 1 <sup>st</sup> Jan 1987–<br>index date | 1 <sup>st</sup> Jan 1987 –<br>31 <sup>st</sup> Dec 2021 |
| Clinical Practice Research<br>Datalink, Aurum (CPRD<br>Aurum) | Clinical Practice Research<br>Datalink (CPRD) | 1 <sup>st</sup> Jan 1995 –<br>index date | 1 <sup>st</sup> Jan 1995 –<br>31 <sup>st</sup> Dec 2021 |
| Hospital Episode Statistics (HES) | Clinical Practice Research<br>Datalink (CPRD) | 1 <sup>st</sup> Jan 1997 – index date | 1 <sup>st</sup> Jan 1997 –<br>31 <sup>st</sup> Dec 2021 |
| Sweden | | | |
| Swedish prescribed drug register (SPDR) <sup>1</sup> | National Board of Health and Welfare | 1 <sup>st</sup> Jul 2005 –<br>index date | 1 <sup>st</sup> Jul 2005 –<br>31 <sup>st</sup> Dec 2020 |
| National patient register (NPR), both inpatient <sup>2</sup> and outpatient <sup>3</sup> registers | National Board of Health and Welfare | Inpatient:<br>1 <sup>st</sup> Jan 1997 –<br>index date | Inpatient:<br>1 <sup>st</sup> Jan 1997 –<br>31 <sup>st</sup> Dec 2020 |
| | | Outpatient:<br>1st Jan 2001 –<br>index date | Outpatient:<br>1 <sup>st</sup> Jan 2001 –<br>31 <sup>st</sup> Dec 2020 |
| Swedish cancer registry (SCR) <sup>4</sup> | National Board of Health and Welfare | 1st Jan 1958 –<br>index date | 1 <sup>st</sup> Jan 1958 –<br>31 <sup>st</sup> Dec 2020 |
| Cause of death register <sup>5</sup> | National Board of Health and Welfare | Not applicable | 1 <sup>st</sup> Jan 2014 – 31 <sup>st</sup> Dec 2020 |
| Total population register <sup>6</sup> | Statistics Sweden | 1st Jan 2013 –<br>index date | 1 <sup>st</sup> Jan 2013 –<br>31 <sup>st</sup> Dec 2020 |
| Longitudinal integration database for health insurance and labor market studies (LISA) <sup>6</sup> | Statistics Sweden | 1 <sup>st</sup> Jan 2013 – index date | 1 <sup>st</sup> Jan 2013 –<br>31 <sup>st</sup> Dec 2020 |
| National diabetes register (NDR) <sup>7</sup> | Centre of Registers,<br>Region Västra Götaland | 1 <sup>st</sup> Jan 2012 – index date | 1 <sup>st</sup> Jan 2012 –<br>31 <sup>st</sup> Dec 2020 |
| Finland | | • | • |

SEAP for non-interventional study BI Study No: 1245.97 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated

| companies | 6 6 | | |
|---|---|---|---|
| Finnish Prescription Register | Social Insurance | 1 <sup>st</sup> Jan 1994 – | 1 <sup>st</sup> Jan 1994 – |
| (FPR) <sup>8</sup> | Institution (SII) | index date | 31st Dec 2020 |
| Finnish Registry for Reimbursed | Social Insurance | 1 <sup>st</sup> Jan 1996 – | 1st Jan 1996 – |
| Medications <sup>9</sup> | Institution (SII) | index date | 31st Dec 2020 |
| Care Register for Health Care | National Institute for | 1 <sup>st</sup> Jan 1996 – | 1st Jan 1996 – |
| (HILMO) <sup>10</sup> | Health and Welfare (THL) | index date | 31st Dec 2020 |
| Register of Primary Health | | 1 <sup>st</sup> Jan 2011 – | 1 <sup>st</sup> Jan 2011 – |
| Care Visits (AvoHILMO) <sup>11</sup> | Health and Welfare (THL) | index date | 31st Dec 2020 |
| Finnish cancer registry (FCR) <sup>12</sup> | Cancer Society of Finland | 1 <sup>st</sup> Jan 1953 – index date | 1 <sup>st</sup> Jan 1953 – 31 <sup>st</sup><br>Dec 2020 |
| Finnish Cause of Death<br>Register <sup>5</sup> | Statistics Finland | Not applicable | 1 <sup>st</sup> Jan 2014 – 31 <sup>st</sup><br>Dec 2020 |
| Four regional EMR databases<br>(Helsinki, Espoo, Vantaa, and<br>Helsinki University Hospital<br>[HUS] area) <sup>6</sup> | Cities of Helsinki, Espoo,<br>and Vantaa, and Helsinki<br>University Hospital | 1 <sup>st</sup> Jan 2013 –<br>index date | 1 <sup>st</sup> Jan 2013 –<br>31 <sup>st</sup> Dec 2020 |
| Population register centre <sup>6</sup> | Population register centre | 1 <sup>st</sup> Jan 2013 – index date | 1 <sup>st</sup> Jan 2013 –<br>31 <sup>st</sup> Dec 2020 |

<sup>&</sup>lt;sup>1</sup> Data since the register was established in July 2005.

## 4.2.4. INCLUSION AND EXCLUSION CRITERIA

The following inclusion/exclusion criteria will be applied to the source population in order to identify the study population in Sweden, Finland and the UK.

Table 2 Inclusion criteria.

| Criteria | Definition | Data source |
|----------|------------|-------------|

<sup>&</sup>lt;sup>2</sup> Data since ICD-10 codes have been used (1997-).

<sup>&</sup>lt;sup>3</sup> Data since the register was established (2001-).

<sup>&</sup>lt;sup>4</sup> Data since the registry was established (1958-).

<sup>&</sup>lt;sup>5</sup> Data since the start of the study period (2014-). However, data will also be extracted since one year before the start of the study period (2013-), as in few cases observations of dispensed study drugs defining the population may occur after death.

<sup>&</sup>lt;sup>6</sup> Data since 1 year before the start of the study period (2013-).

<sup>&</sup>lt;sup>7</sup> Data since 2 years before the start of the study period (2012-).

<sup>&</sup>lt;sup>8</sup> Data since the register was established (1994-).

<sup>&</sup>lt;sup>9</sup> Data since the register was established (1996-).

<sup>&</sup>lt;sup>10</sup> Data since ICD-10 codes have been used (1996-).

<sup>&</sup>lt;sup>11</sup> Data since the register was established (2011-).

<sup>&</sup>lt;sup>12</sup> Data since the register was established (1953-).

| Diagnosis of type 2 diabetes | A diagnosis of type 2-diabetes mellitus (T2DM) identified using the country-specific | UK: CPRD-GOLD and Aurum |
|---|---|---|
| | algorithms detailed below. | Sweden: NDR, National |
| | ATC codes are provided in Annex II. | Patient Register (NPR), and SPDR |
| | | Finland: avoHILMO, FPR, and |
| | All available data prior to index date <sup>2</sup> inclusive. | Reimbursement register |
| Age over 18 years at | Patient age over 18 years. | UK: CPRD-GOLD and |
| index date | Evaluated at index date <sup>2</sup> . | Aurum |
| | | Sweden: SPDR |
| | | Finland: FPR and<br>Population register<br>centre |
| At least one year of database membership | Difference between index date and database membership start $\geq$ 365 days. | UK: CPRD-GOLD and Aurum |
| | Evaluated at index date <sup>2</sup> | Sweden: Total population register <sup>1</sup> |
| | | Finland Population register centre |
| Inclusion criteria verified | All of the above. | |

The national patient register will be used if data on immigration/emigration are unavailable from the Total population register.

The following country-specific algorithms will be used for the identification of a diagnosis of T2DM at or prior to index date date:

#### UK

A diagnosis of T2DM will be identified using relevant diagnosis codes (listed in Annex I) in CPRD-GOLD (clinical and therapy data) or CPRD Aurum (observation and problem data).

#### **Sweden**

Patients with a diagnosis of T2DM will be identified in following steps:

- Search for a diagnosis of T2DM in NDR data (diabetes registry records) using the corresponding variables that indicate the registered type of diabetes.

<sup>&</sup>lt;sup>2</sup> The index date is defined as the date of first purchase/prescription of empagliflozin or a DPP-4 inhibitor during the study period (from August 1, 2014 until December 31, 2020, 2021 for CPRD).

- If no T2DM diagnosis is present in NDR data, search for a diagnosis in NPR data (inpatient and outpatient records) using the relevant ICD-10 diagnosis codes listed in Annex I.
- If no T2DM diagnosis is present in NDR or NPR, search for a previous (before index date) prescription of metformin in SPDR data using the ATC codes listed in Annex II.

#### **Finland**

Patients with a diagnosis of T2DM will be identified in following steps:

- Search for a diagnosis of T2DM in the reimbursement register using ICD-10 diagnosis codes listed in Annex I.
- If no T2DM diagnosis is present in the reimbursement register, search for a main diagnosis in AvoHILMO data using relevant ICD-10 diagnosis codes listed in Annex I.
- If no T2DM diagnosis is found in the reimbursement register or in AvoHILMO, search for a previous (before index date) prescription of metformin using the ATC codes listed in Annex II.

#### **Exclusion criteria**

Table 3 Exclusion criteria.

| Criteria | Definition | Data source |
|---|---|---|
| History of cancer prior to index date | A registered diagnosis of any cancer (excluding non-melanoma skin cancer) | UK: CPRD-GOLD and Aurum |
| | (ICD-10, ICD-7, ICD-O-3 and READ diagnosis codes in Annex I) | Sweden: Swedish cancer registry (SCR) |
| | All available medical history prior to index date inclusive. | Finland: Finnish cancer registry (FCR) |
| Diabetes diagnosis other than type 2 | A diagnosis of type 1 diabetes mellitus (T1DM) or other non-type 2 diabetes | UK: CPRD-GOLD and Aurum |
| | identified using the country-specific identification algorithms described below. | Sweden: NDR and NPR |
| | Relevant ICD-10 codes and READ diagnosis codes are provided in Annex I. | Finland: Reimbursment registry |
| | All available medical history prior to index date inclusive. | |

SEAP for non-interventional study BI Study No: 1245.97

| companies | | |
|---|---|---|
| SGLT-2 inhibitor or DPP-4 inhibitor use any | Any prescription of a SGLT-2 inhibitor drug (including empagliflozin) or a DPP-4 | UK: CPRD-GOLD and Aurum |
| time prior to index date | inhibitor drug, alone or in combination. | Sweden: SPDR |
| | (ATC codes in Annex II) | Finland: FPR |
| | All available prescription history prior to index date exclusive. | |
| combinations of SGLT- | Any prescription record of a SGLT-2 inhibitor drug in combination with a DPP- | UK: CPRD-GOLD and Aurum |
| 2 inhibitors with DPP-4 inhibitors or | 4 inhibitor drug. | Sweden: SPDR |
| empaglifozin. | (ATC codes in Annex II) | Finland: FPR |
| . 0 | All available prescription history prior to index date inclusive. | |
| End-stage renal disease diagnosis or receipt of | Any registered record with a diagnosis or procedures of end-stage renal disease, | UK: CPRD-GOLD and Aurum |
| renal dialysis any time prior to index date | receipt of renal dialysis or eGFR $\leq 15$ (ml/min/1.73 m <sup>2</sup> ). | Sweden: NPR and NDR |
| | (ICD-10 codes, procedure codes and READ diagnosis codes in Annex I) | Finland: HILMO and AvoHILMO |
| | All available medical history prior to index date inclusive. | |
| Patient excluded from the study population | Any of the above exclusion criteria verified prior to enrolment. | |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated

The following country-specific algorithms will be used to identify patients with a diagnosis of any diabetes other than T2DM for exclusion criteria:

#### UK

Patients with a diagnosis of any diabetes other than T2DM will be identified in CPRD-GOLD (clinical and therapy data) or CPRD Aurum (observation and problem data) using relevant diagnosis codes (listed in Annex I).

#### Sweden

Patients with a diagnosis of any diabetes other than T2DM will be identified in following steps:

- Search for a diagnosis of any diabetes other than T2DM in NDR data using the corresponding variables that indicate the registered type of diabetes.
- For patients without a diagnosis of diabetes other than T2DM in NDR, search for a main diagnosis of T1DM in NPR data (inpatient and outpatient records) using the

relevant ICD-10 diagnosis codes listed in Annex I. A T1DM diagnosis will be confirmed and the patient is excluded if the latest event with a main diagnosis of T1DM is not succeeded by an event with a main diagnosis of T2DM within the look-back period.

#### **Finland**

Patients with a diagnosis of any diabetes other than T2DM will be identified in the reimbursement register using relevant ICD-10 diagnosis codes listed in Annex I.

#### 5. VARIABLES

#### 5.1. EXPOSURES

#### **5.1.1. STUDY MEDICATIONS**

#### **Main Cohort:**

In each country, after identifying the study cohort, patients will be grouped in two exposure groups:

- New users of empagliflozin: Patients prescribed empagliflozin at index date.
- New users of DPP-4 inhibitors: Patients prescribed any DPP-4 inhibitor at index date.

## Sub-cohort of users of empagliflozin in combination with metformin

Patients using metformin in free or fixed dose combination will be identified in the main study cohort and grouped in two exposure groups for a separate analysis:

- Patients prescribed empagliflozin in free or fixed dose combination with metformin at index date.
- Patients prescribed any DPP-4 inhibitor in free or fixed dose combination with metformin at index date.

#### **5.1.2. INDEX DATE**

The index date is defined as the date of first dispensation/prescription of empagliflozin or of a DPP-4 inhibitor during the study period (from 1st August, 2014 until 31st December, 2020 – 2021 for UK-CPRD).

#### **5.1.3. EXPOSURE TIME**

Time at risk will start on index date and continue until first treatment discontinuation (see definition in Section 5.1.6). Continuous exposure will be defined as successive exposure periods for the study drugs separated by gaps of 30 days at most. Duration of exposure

episodes for individual prescriptions of study drugs will be derived based on package size, unit strength and daily dose.

To account for an empirical induction/promotion period of cancer, a latency period of 6 months (180 days) after the index date is applied. Patients with less than 6 months (180 days) of follow-up time will be excluded. In addition, patients with any diagnosis of any cancer within the latency period will be excluded. In a sensitivity analysis, the latency period will be extended to 12 months (365 days).



<sup>\*</sup> Other drugs: a prescription of another drug (empagliflozin, a DPP-4 inhibitor, or a SGLT-2 inhibitor) other than index drug

Figure 1 Definition of continous exposure period of index drug

For the primary AT analyses, the time at risk will begin after the latency period and end at urinary tract (bladder, renal or other) cancer or at any of the censoring events (listed in Table 4), whichever occurs first. In addition, treatment discontinuation of the index drug (defined in Section 5.1.6) is an additional censoring variable.

For the sensitivity ITT analyses, the time at risk will begin after the latency period and end at urinary tract (bladder, renal or other) cancer or any of the censoring events excluding treatment discontinuation of the index drug.

Patients with censored time at risk will not be able to re-enter the study cohort at a later time point. The time at risk will not be censored if oral or injectable glucose-lowering drugs other than the index drugs and SGLT-2 inhibitors are prescribed in addition to empagliflozin or a DPP-4 inhibitor after the index date.

Table 4 Censoring events.

| Censoring event | Definition | Data source |
|---|---|---|
| All-cause mortality | Censoring of follow-up time occurs at the date of death regardless of the cause. | UK: CPRD-GOLD and Aurum |
| | Applied in all analyses. | Sweden: Cause of death register |
| | | Finland: Cause of death register |
| Emigration from the study country | Censoring of follow-up time occurs at the date of emigration from the study country. | UK: CPRD-GOLD and Aurum |
| | Applied in all analyses. | Sweden: Total population register <sup>1</sup> |
| | | Finland: Population register centre |
| Patient transfer | Censoring of follow-up time occurs at the date of patient transfer. | UK: CPRD-GOLD and Aurum |
| | Applied in all analyses. | Sweden: NA |
| | | Finland: NA |
| Incidence of any cancer during follow-up | A registered diagnosis of any cancer (excluding non-melanoma skin cancer) | UK: CPRD-GOLD and Aurum |
| | during follow-up. (ICD-10, ICD-7, ICD-O-3 and READ | Sweden: Swedish cancer registry (SCR) |
| | diagnosis codes in Annex I) | Finland: FCR |
| | Applied in all analyses. | |
| Diabetes diagnosis other than type 2 | A diagnosis of type 1 diabetes or other<br>non-type 2 diabetes during follow-up<br>identified using the same algorithm as<br>used for the exclusion criteria (Section<br>4.2.4) | UK: CPRD and Aurum Sweden: NDR, NPR Finland: reimbursement |
| | Relevant ICD-10 codes and READ diagnosis codes are provided in Annex I. | registry |
| | Applied in all analyses. | |
| End of study period | Censoring of follow-up time occurs at end of study date i.e. 31 December 2020 (2021 for UK-CPRD). | NA |
| | Applied in all analyses. | |

| Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | |
|---|---|---|
| Treatment discontinuation (AT exposure- main analysis) | Censoring of follow-up time occurs 90 days after - last day of medication (i.e. stop date) - new prescription of the other study drug or of a SGLT-2 inhibitor Applied only in analyses using the AT exposure definition. | UK: CPRD-GOLD and<br>Aurum Sweden: SPDR Finland: FPR |
| Treatment discontinuation (AT exposure- sensitivity analysis) | Censoring of follow-up time occurs 180 days after - last day of medication (i.e. stop date) - new prescription of the other study drug or of a SGLT-2 inhibitor Applied only in the sensitivity analysis using the AT exposure definition. | UK: CPRD-GOLD and<br>Aurum<br>Sweden: SPDR<br>Finland: FPR |

<sup>&</sup>lt;sup>1</sup> The National patient register will be used if data on immigration/emigration are unavailable from the Total population register.

# 5.1.4. Days' supply and duration of exposure

The estimated days' supply of each prescription/dispensing will be used to determine exposure episodes. Continuous exposure periods will then consist of consecutive exposure episodes separated by a gap of at most 30 days (Section 5.1.6).

The construction of exposure episodes is based on the assumptions that the total prescribed/dispensed dose is consumed as 1 unit per day, 1 defined daily dosage (DDD) per day, or 1 prescribed daily dose (PDD) per day. The construction of exposure episodes using PDD exihibited better performance and led to fewer outcome misclassifications, compared to the alternative approaches [4]. In this study, the length of each exposure episode (days' supply) will be calculated at the prescription level as the total prescribed/dispensed doses divided by the daily dose.

The total doses will be calculated as the total number of product units per prescription, using corresponding variables including the package size, unit strength and prescribed number of packages. The daily dose in product units will be determined based on the PDD (or recommended daily dose) and the unit strength in the prescribed packages. For study drugs, the daily doses will be ascertained from recommended dosages and pill strength. In case of missing information, the days' supply will be estimated as the median days' supply of the same drug prescription. The available variables will be extracted from the relevant databases, as described below.

SEAP for non-interventional study BI Study No: 1245.97

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **UK CPRD-GOLD and Aurum**

The total doses will be estimated as the total number of prescribed units using the follow variables provided by CPRD:

- Number of individual product packs prescribed
- Pack size
- Unit strength of the product

For study drugs and metformin, daily dose and days' supply will be derived from pill strength and dosage recommendations. For other drugs, the daily dose will be ascertained based on the prescribed daily dose (if available) or defined daily dose and the unit strength of the dispensed packages.

#### Sweden

The total doses will be calculated as the total number of dispensed units using the follow variables:

- Size of dispensed package
- Number of dispensed packages
- Drug strength

For study drugs and metformin, daily dose and days' supply will be derived from pill strength and dosage recommendations as described in Annex IV. For other drugs, the daily dose will be ascertained based on the defined daily dose and the unit strength of the dispensed packages.

#### **Finland**

The prescription information are available as purchase records, including

- ATC codes
- Number of packages prescribed
- Nordic Article Number (VNR).

VNRs will be mapped to retrieve information on the package size and unit strength of the products, using the publically available database from Finnish Medicines Agency (FIMEA). For study drugs and metformin, daily dose and days' supply will be derived from pill strength and dosage recommendations as described in Annex IV. For other drugs, the daily dose will be ascertained based on the defined daily dose and the unit strength of the dispensed packages.

#### **5.1.5.** Dose

Dose will be the current daily dose as described in Table 6.

The current daily dose will be derived from pill strength and dosage recommendations as described in Section 5.1.5.

#### 5.1.6. Definition of continuous treatment and discontinuation

#### **Continuous treatment**

Continuous treatment is defined as having consecutive treatment episodes separated by a grace period of 30 days (Figure 1). In a sensitivity analysis, the grace period is extended to 90 days.

In case of overlaps between treatment episodes (i.e., a new prescription/dispensation during an ongoing exposure period), the overlapping days are added to the end of the following treatment episode, resulting in a longer treatment episode to take into account possible stockpiling.

#### **Treatment discontinuation**

Treatment discontinuation (see Table 4) is defined either by

- The start of a new prescription of any new drug from the following drug groups: empagliflozin, DPP-4 inhibitors, or SGLT-2 inhibitors), or of a fixed-dose combination of a SGLT-2 inhibitor with a DPP-4 inhibitor (identified from the ATC class A10BD)
- The end date of the first continuous exposure period of the index drug (stop date) plus a 3-month (90 days) period following it.

The discontinuation date is defined as the stop date/start date of a new drug plus 90 days.

## 5.1.7. Primary Exposure definition

The primary definition of exposure, i.e. as-treated exposure (AT), is defined as a continuous exposure to empagliflozin or to a DPP-4 inhibitor, starting from index date. Continuous exposure and treatment discontinuation are defined in Section 5.1.6.

In the Swedish dataset, drug exposure will be identified from SPDR. In Finland, the FPR will be used. In the UK datasets, drug exposure will be identified from CPRD data. The study drugs will be identified using ATC codes (med codes for CPRD) listed in Annex II.

Table 5 As-treated exposure definition

| Exposure | Definition | Details | Data source |
|---|---|---|---|
| Exposure to index drugs (as treated) | Exposure status for empagliflozin (alone or in combination with metformin) or DPP-4 inhibitor (including | Time-fixed Categorical: | UK: CPRD Sweden: SPDR |
| | combinations) based on purchased amounts and daily defined dose. | Empagliflozin DPP-4 inhibitor | Finland: FPR |
| | ATC codes for empagliflozin and DPP-4 inhibitors in Annex II. | | |
| | Evaluated at index date | | |

# 5.1.8. SECONDARY EXPOSURE DEFINTIONS

# Exposure definitions based on dosage or duration

Table 6 Exposure definitions based on dosage or duration

| Exposure | Definition | Details | Data source |
|---|---|---|---|
| Cumulative dose of | a empadiflazin dase consumption based | Time-dependent | UK: CPRD |
| empagliflozin use in grams | | Categorical <sup>1</sup> : | Sweden: SPDR |
| Similia | purchased amounts since the start of | Never | Finland: FPR |
| | follow-up. ATC codes for empagliflozin in | 0 - <cumulative dose="" q1<="" td=""><td></td></cumulative> | |
| | Annex II. | | |
| | Updating from index date onwards.* | $\geq$ Q2 to $\leq$ Q3 | |
| | | ≥ Q3 | |
| Daily dose of | The dosage of empagliflozin prescribed | Time-dependent | UK: CPRD |
| empagliflozin | per daily use (10mg vs. 25mg). | Categorical: | Sweden: SPDR |
| | ATC codes for empagliflozin in Annex II. | Never | Finland: FPR |
| | Updating from index date onwards.* | 10 mg | |
| | | 25 mg | |

| Cumulative exposure duration to empagliflozin in months | Time-updating cumulative sum of duration since the first use of empagliflozin (alone or in combination with metformin), in months. | Time-dependent<br>Categorical <sup>2</sup> :<br>Never | UK: CPRD<br>Sweden: SPDR<br>Finland: FPR |
|---|---|---|---|
| | ATC codes for empagliflozin in Annex II. | 0 - < cumulative duration Q1 | |
| | Updating from index date onwards.* | $\geq$ Q1 to $\leq$ Q2 | |
| | | $\geq$ Q2 to $<$ Q3 | |
| | | $\geq$ Q3 | |

<sup>\*</sup>The last observed value will be carried forward for 3 months (90 days) to account for the 90-day delay between end of treatment and treatment discontinuation as defined in Section 5.1.6.

## Intention-to-treat exposure definition

The intention to treat exposure definition assumes that individuals do not discontinue the treatment of an index drug.

Table 7 Intention-to-treat exposure definition

| Exposure | Definition | Details | Data source |
|---|---|---|---|
| Exposure to index drugs (Intention to treat) | Purchase of empagliflozin (alone or in combination with metformin) or any DPP-4 inhibitors (including combinations). | Time-fixed | UK: CPRD |
| | | Categorical: | Sweden: SPDR |
| | | Empagliflozin | Finland: FPR |
| | ATC codes for empagliflozin and DPP-4 inhibitors in Annex II. | DPP-4 inhibitor | |
| | Evaluated at index date. | | |

## 5.2. OUTCOMES

#### **5.2.1. Primary outcomes**

The outcomes of interest for this study are urinary tract cancers, bladder cancer, and renal cancer. These outcomes will be identified through Clinical Practice Research Datalink's General Practitioner OnLine Data (CPRD-GOLD and CPRD Aurum) data in the UK, the Swedish cancer registry (SCR) in Sweden and Finnish cancer registry (FCR) in Finland.

<sup>&</sup>lt;sup>1</sup> The categories are defined based on the quartiles of overall cumulative dose (grams) of the study population

<sup>&</sup>lt;sup>2</sup> The categories are defined based on the quartiles of overall cumulative exposure duration (months) of the study population

Table 8 Main outcomes

| Outcome | Definition | Details | Data source |
|---|---|---|---|
| Urinary tract cancer (malignant or carcinoma in situ) | First record of urinary tract cancer (ICD-10, ICD-O-3 and READ diagnosis codes in Annex I). | Time to first event during follow-up. | UK: CPRD-<br>GOLD and<br>Aurum |
| | During follow-up. | | Sweden: SCR |
| | | | Finland: FCR |
| Bladder cancer<br>(malignant and<br>carcinoma in<br>situ) | First record of bladder cancer (ICD-10, ICD-O-3 and READ diagnosis codes in Annex I). <b>During follow-up.</b> | Time to first event during follow-up. | UK: CPRD-<br>GOLD and<br>Aurum |
| | Dailing Tollow up. | | Sweden: SCR |
| | | | Finland: FCR |
| Renal cancer (malignant) | First record of renal cancer (ICD-10, ICD-O-3 and READ diagnosis codes in Annex I). <b>During follow-up.</b> | Time to first event during follow-up. | UK: CPRD-<br>GOLD and |
| | | | Aurum |
| | | | Sweden: SCR |
| | | | Finland: FCR |

The date of diagnosis of the first incidence of urinary tract cancers as specified in CPRD-GOLD and CPRD Aurum, in the SCR or in the FCR after the entry into the study will be used as the primary outcome date.

In the Swedish and Finnish datasets, urinary tract cancer events will be identified from the SCR and FCR using ICD-10 and ICD-O-3 codes (Annex I). In CPRD, urinary tract cancer events will be identified in CPRD-GOLD using READ codes and in CPRD Aurum using READ and

SNOMED CT codes (Annex I).



# **5.3. COVARIATES**

# 5.3.1. Demographics and other baseline variables

Table 11 Demographics and other baseline variables.

| Variable | Definition | Details | Data source |
|---|---|---|---|
| Age at index | Patient age at index. | Time-fixed | UK: CPRD |
| | Evaluated at index date. | Continuous<br>Categorical:<br>18-49<br>50-64<br>65-69<br>70-74<br>75-79<br>80-84<br>85 and over | Sweden: SPDR<br>Finland: FPR,<br>Population<br>register centre |
| Sex | Patient sex. Evaluated at index date. | Time-fixed Categorical: Female Male | UK: CPRD Sweden: SPDR Finland: Population register centre |
| Highest level of education | Patient highest level of education Evaluated for the calendar year of the index date. | Time-fixed Categorical: Compulsory Upper secondary Post secondary | UK: N/A Sweden: Longitudinal integration database for health insurance and labor market studies (LISA) Finland: Statistics Finland |

| Disposable income, individual at index | Patient available income. | Time-fixed | UK: N/A |
|---|---|---|---|
| | Evaluated for the calendar year of the index date. | Categorical: <sup>1</sup> | Sweden: LISA<br>Finland: N/A |
| | | < Q1 | |
| | | $\geq$ Q1 $-<$ Q2 | |
| | | $\geq$ Q2 $ <$ Q3 | |
| | | $\geq$ Q3 | |
| Disposable | Patient family income. | Time-fixed | UK: N/A |
| income, family at index | <b>Evaluated for the calendar year of the index date.</b> | Continuous<br>Categorical: <sup>1</sup> | Sweden: LISA<br>Finland: N/A |
| | | < Q1 | |
| | | $\geq$ Q1 $-<$ Q2 | |
| | | $\geq$ Q2 $-<$ Q3 | |
| | | $\geq$ Q3 | |
| Socioeconomic | Socioeconomic status based on area of | Time-fixed | UK: CPRD |
| summary<br>variable | residence. | Categorical: | Sweden: N/A |
| variable | Evaluated at index date. | | Finland: N/A |
| CPRD database | Source of CPRD data | Time-fixed | UK: CPRD |
| | Evaluated at index date. | Categorical: | Sweden: N/A |
| | | GOLD | Finland: N/A |
| | | Aurum | |
| • | Calendar year of index date. | Time-fixed | UK: CPRD |
| index date | Evaluated at index date. | Categorical: | Sweden: SPDR |
| | | 2014 | Finland: FPR |
| | | 2015 | |
| | | 2016 | |
| | | 2017 | |
| | | 2018 | |
| | | 2019 | |
| | | 2020 | |
| | | 2021 | |
SEAP for non-interventional study BI Study No: 1245.97

| Duration of | Time difference between index date and | Time-fixed | UK: CPRD |
|---|---|---|---|
| look-back period<br>(in years) | database membership start. Evaluated at index date. | Continuous Categorical: | Sweden: Total population register <sup>2</sup> |
| | | 2-5<br>6-9 | Finland: Population register centre |
| | | 10 and over | register centre |
| BMI | Patient BMI value at index. | Time-fixed | UK: CPRD |
| | Evaluated at index date using closest value. | Continuous<br>Categorical: <sup>2</sup> | Sweden: NDR<br>Finland: |
| | | <20 | AvoHILMO, |
| | | ≥20-24.9 | EMR |
| | | 25-29.9 | databases |
| | | >30 | |
| Smoking status | Patient smoking status at index date. | Time-fixed | UK: CPRD |
| | Evaluated at index date using closest value. | Categorical: | Sweden: NDR |
| | | $Yes^3$ | Finland: |
| | | No | AvoHILMO,<br>EMR<br>databases |
| Alcohol use | Patient alcohol use status at index date. | Time-fixed | UK: CPRD |
| status | Evaluated at index date using closest value. | Categorical: | Sweden: NA |
| | | Yes | Finland: NA |
| | | No | |
| HbA1c value (in mmol/mol) | Time-dependent HbA1c measurement value in mmol/mol. | Time-<br>dependent | UK: CPRD<br>Sweden: NDR |
| | Initialized at index using closest value to index date and updating from index date | Continuous Categorical: | Finland: EMR databases |
| | onwards. | < 48 (6.5%) | |
| | | ≥48 (6.5 %)-<br><64 (8 %) | |
| | | ≥64 (8%) | |

| Number of | The number of albuminuria tests received by | Time-fixed | UK: CPRD |
|---|---|---|---|
| albuminuria tests | the patient prior to index date. | Continuous | Sweden: NDR |
| | Evaluate at index using all available history prior to index date. | | Finland: EMR databases |

# 5.3.2. Concomitant diseases

Table 12 Diabetic complications variables.

| Variable | Definition | Details | Data source |
|---|---|---|---|
| Time since first<br>diabetes<br>diagnosis at<br>index date | Time difference between [index date] and [first type 2 diabetes diagnosis date]. ICD-10 and READ diagnosis codes for type 2 diabetes in Annex I. Evaluated at index date. | Time-fixed Continuous Categorical: < Q1 ≥ Q1-< Q2 ≥ Q2-< Q3 ≥ Q4 | UK: CPRD<br>Sweden: NDR<br>Finland: HILMO,<br>AvoHILMO |
| Duration of treated diabetes at index date | Time difference between [index date] and [first antidiabetic treatment prescription/purchase date] in the data. ATC codes for antidiabetic treatment in Annex II. Evaluated at index date. | Time-fixed<br>Continuous | UK: CPRD Sweden: SPDR Finland: FPR |
| Diabetic complications at index date | The variable is evaluated at index date and indicates the number of recorded diagnoses of diabetic complications using all available history prior to index date. ICD-10, READ diagnosis codes and corresponding NDR variables for diabetic complications in Annex I. Evaluated at index using all available history prior to index date. | Time-fixed Continous Categorical: 0 1-2 >2 | UK: CPRD<br>Sweden: NPR<br>NDR<br>Finland: HILMO,<br>AvoHILMO |

The national patient register will be used if data on immigration/emigration are unavailable from the Total population register.

Categories under-weight (<20), normal weight (20-24.9), overweight (25-29.9), and obese (>30) may be adjusted based on the observed

distribution of the data.

<sup>3</sup> In Sweden, a smoker is a patient smoking one or more cigarettes per day or a pipe daily or who had stopped smoking within the past 3 months. If data allows, categories current, never, past will be used.

SEAP for non-interventional study BI Study No: 1245.97

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or on

| ne variable is evaluated at index date and | Time-fixed | UK: CPRD |
|---|---|---|
| dicates a register record with a diagnosis of abetic retinopathy or diabetic maculopathy ing all available history prior to index date. | Categorical:<br>Yes | Sweden: NPR NDR |
| CD-10, READ diagnosis codes and orresponding NDR variables for diabetic tinopathy or diabetic maculopathy in nnex I. | No | Finland: HILMO,<br>AvoHILMO |
| valuated at index using all available story prior to index date. | | |
| ne variable is evaluated at index date and | Time-fixed | UK: CPRD |
| | Categorical: | Sweden: NPR |
| ior to index date. | Yes | Finland: HILMO, |
| D-10 and READ diagnosis codes for abetic nephropathy in Annex I. | No | AvoHILMO |
| valuated at index using all available story prior to index date. | | |
| ne variable is evaluated at index date and | Time-fixed | UK: CPRD |
| indicates a register record with a diagnosis of diabetic neuropathy using all available history | Categorical:<br>Yes | Sweden: NPR<br>Finland: HILMO, |
| D-10 and READ diagnosis codes for abetic neuropathy in Annex I. | No | AvoHILMO |
| valuated at index using all available story prior to index date. | | |
| ne variable is evaluated at index date and | Time-fixed | UK: CPRD |
| | Categorical: | Sweden: NPR |
| story prior to index date. | Yes | Finland: HILMO, |
| CD-10 and READ diagnosis codes for eripheral vascular disease in Annex I. | No | AvoHILMO |
| valuated at index using all available story prior to index date. | | |
| | ing all available history prior to index date. D-10, READ diagnosis codes and presponding NDR variables for diabetic inopathy or diabetic maculopathy in innex I. In aluated at index using all available story prior to index date. The variable is evaluated at index date and dicates a register record with a diagnosis of abetic nephropathy using all available history or to index date. D-10 and READ diagnosis codes for abetic nephropathy in Annex I. The variable is evaluated at index date and dicates a register record with a diagnosis of abetic neuropathy using all available story prior to index date. The variable is evaluated at index date and dicates a register record with a diagnosis of abetic neuropathy using all available history or to index date. D-10 and READ diagnosis codes for abetic neuropathy in Annex I. The valuated at index using all available story prior to index date. The variable is evaluated at index date and dicates a register record with a diagnosis of ripheral vascular disease using all available story prior to index date. D-10 and READ diagnosis codes for ripheral vascular disease in Annex I. The valuated at index using all available at or prior to index date. D-10 and READ diagnosis codes for ripheral vascular disease in Annex I. The valuated at index using all available at or prior to index date. | politic retinopathy of diabetic maculopathy ing all available history prior to index date. D-10, READ diagnosis codes and presponding NDR variables for diabetic inopathy or diabetic maculopathy in innex I. Taluated at index using all available story prior to index date. Time-fixed Categorical: Yes D-10 and READ diagnosis codes for abetic nephropathy in Annex I. Taluated at index using all available story prior to index date. Time-fixed Categorical: Yes No Time-fixed Categorical: Yes Time-fixed Categorical: Yes No No Time-fixed Categorical: Yes No |

SEAP for non-interventional study BI Study No: 1245.97 

| Diabetic lower<br>limb severe<br>complications at<br>index date | The variable is initialized at index date and indicates a register record with a diagnosis of diabetic lower limb severe complications using all available history prior to index date. | Time-fixed Categorical: Yes | UK: CPRD Sweden: NPR Finland: HILMO, |
|---|---|---|---|
| | ICD-10 and READ diagnosis codes for diabetic lower limb severe complications in Annex I. | No | AvoHILMO |
| | Evaluated at index using all available history prior to index date. | | |

<sup>&</sup>lt;sup>1</sup> Categories to be defined based on the observed distribution of the data.

Table 13 Other non-diabetic concomitant disease variables.

| Variable | Definition | Details | Data source |
|---|---|---|---|
| Kidney or genitourinary stones | nitourinary indicates a register record with a diagnosis of Categorical: | Yes | UK: CPRD Sweden: NPR Finland: HILMO, AvoHILMO |
| | Initialized at index and updating from index date onwards. | | |
| Estimated glomerular filtration rate (eGFR) at index date | eGFR estimate derived from serum creatinine measurement using the CKD-Epi equation: eGFR (mL/min/1.73 m²) = 141 x min(S <sub>cr</sub> /K,1)³ x max(S <sub>cr</sub> /K,1)¹-1.209 x 0.993 <sup>Age</sup> x 1.018 [if female]. a = -0.329 (females) or -0.411 (males). Evaluated at index using closest value to index date. | Time-fixed Continuous Categorical <15 (ml/min/1.73 m2) (kidney failure) 15-29 (ml/min/1.73 m2) (severely decreased) 30-44 (ml/min/1.73 m2) (Moderately to severely decreased) 45-59 (ml/min/1.73 m2) (Mildly to moderately decreased) 60-89 (ml/min/1.73 m2) (Mildly decreased) ≥90 (ml/min/1.73 m2) (Mildly decreased) ≥90 (ml/min/1.73 m2) (Normal) | UK: CPRD Sweden: NDR Finland: EMR databases |

SEAP for non-interventional study BI Study No: 1245.97

| <del></del> | | | cpp.p |
|---|---|---|---|
| Renal impairment at index date | The variable is evaluated at index date and indicates an eGFR < 60 (ml/min/1.73 m2) in all available history prior to index date. | Time-fixed | UK: CPRD |
| | | Categorical | Sweden: NDR |
| | Evaluated at index date using all available | Yes | Finland: EMR databases |
| | history prior to index date. | No | uatavases |
| UTI or | The variable is initialized at index date and | Time-dependent | UK: CPRD |
| pyelonephritis | indicates a register record with a diagnosis of UTI or pyelonephritis using all available | Categorical: | Sweden: NPR |
| | history. If no diagnosis prior to index date, it is | Yes | Finland: |
| | time-updated to indicate any diagnosis of UTI | No | HILMO, |
| | or pyelonephritis after index date. | | AvoHILMO |
| | ICD-10 and READ diagnosis codes for UTI or pyelonephritis in Annex I. | | |
| | Initialized at index and updating from index | | |
| | date onwards. | | |
| Liver disease at | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
| index date | indicates a register record with a diagnosis of liver disease using all available history prior to index date. ICD-10 and READ diagnosis codes for liver | Categorical: | Sweden: NPR |
| | | Yes | Finland: |
| | | No | HILMO, |
| | disease in Annex I. | | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |
| ICU admission | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
| at index date | indicates a record of ICU admission in all available history prior to index date. | Categorical: | Sweden: NA |
| | Evaluated at index date using all available | Yes | Finland:<br>HILMO, |
| | history prior to index date. | No | AvoHILMO |
| Pancreatitis at index date | The variable is evaluated at index date and indicates a register record with a diagnosis of | Time-fixed | UK: CPRD |
| | pancreatitis using all available history prior to | Categorical: | Sweden: NPR |
| | index date. | Yes | Finland:<br>HILMO, |
| | ICD-10 and READ diagnosis codes for pancreatitis in Annex I. | No | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |

SEAP for non-interventional study BI Study No: 1245.97 

| Congestive heart failure at index date | The variable is evaluated at index date and indicates a register record with a diagnosis of congestive heart failure using all available | Time-fixed | UK: CPRD |
|---|---|---|---|
| | | Categorical: | Sweden: NPR |
| | history prior to index date. | Yes | Finland: |
| | ICD-10 and READ diagnosis codes for | No | HILMO, |
| | congestive heart failure in Annex I. | | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |
| Systolic blood | Systolic blood pressure measurement value in | Time-fixed | UK: CPRD |
| pressure at index date | mm Hg at index date. | Continuous | Sweden: NDR |
| date | Evaluated at index using closest value to index date. | Categorical <sup>1</sup> : | Finland: EMR |
| | muca uate. | < 120 | databases |
| | | ≥120-<139 | |
| | | ≥140-<159 | |
| | | ≥160 | |
| Diastolic blood | Diastolic blood pressure measurement value in | Time-fixed | UK: CPRD |
| pressure at index date | mm Hg at index date. | Continuous | Sweden: NDR |
| date | index date. | Categorical: <sup>2</sup> | Finland: EMR databases |
| | | < 80 | |
| | | ≥80-89 | |
| | | ≥90-99 | |
| | | 100 or higher | |
| Hypertension at | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
| index date | indicates a register record with a diagnosis of hypertension, or two records within 6 months | Categorical: <sup>2</sup> | Sweden: NPR, |
| | (180 days) of systolic blood pressure $\geq$ 140 and | Yes | NDR |
| | diastolic blood pressure $\geq 90$ using all available history prior to index date. | No | Finland: HILMO, |
| | ICD-10 and READ diagnosis codes for | | AvoHILMO, |
| | hypertension in Annex I. | | EMR databases |
| | Evaluated at index date using all available history prior to index date. | | |

| Stroke at index | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
|---|---|---|---|
| date | indicates a register record with a diagnosis of<br>stroke using all available history prior to index | Categorical: | Sweden: NPR |
| | date. | Yes | Finland:<br>HILMO, |
| | ICD-10 and READ diagnosis codes for stroke in Annex 1. | No | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |
| Myocardial | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
| infarction at index date | indicates a register record with a diagnosis of myocardial infarction using all available | Categorical: | Sweden: NPR |
| macx date | history prior to index date. | Yes | Finland: |
| | ICD-10 and READ diagnosis codes for | No | HILMO, |
| | myocardial infarction in Annex I. | | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |
| Autoimmune | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
| disease at index date | indicates a register record with a diagnosis of<br>autoimmune disease using all available history<br>prior to index date. | Categorical: | Sweden: NPR |
| date | | Yes | Finland: |
| | ICD-10 and READ diagnosis codes for | No | HILMO, |
| | autoimmune disease in Annex I. | | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |
| COPD at index | The variable is evaluated at index date and | Time-fixed | UK: CPRD |
| date | indicates a register record with a diagnosis of COPD using all available history prior to index | Categorical: | Sweden: NPR |
| | date. | Yes | Finland: |
| | ICD-10 and READ diagnosis codes for COPD | No | HILMO, |
| | in Annex I. | | AvoHILMO |
| | Evaluated at index date using all available history prior to index date. | | |

<sup>&</sup>lt;sup>1</sup> Modification of Diet in Renal Disease (MDRD) study <a href="http://clinchem.aaccjnls.org/content/53/4/766.long">http://clinchem.aaccjnls.org/content/53/4/766.long</a>

 $<sup>^2\,</sup>http://www.heart.org/HEARTORG/Conditions/HighBloodPressure/AboutHighBloodPressure/Understanding-Blood-Pressure-Readings\_UCM\_301764\_Article.jsp\#$ 

SEAP for non-interventional study BI Study No: 1245.97

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5.3.3. Concomitant medications

Table 14 Other diabetic medication exposure definitions

| Exposure | Definition | Details | Data source |
|---|---|---|---|
| Concomitant | Variable indicating the concomitant use of | Time-fixed | UK: CPRD |
| use of insulin at index date | , , , | Categorical: | Sweden: SPDR |
| | | Yes | Finland: FPR |
| | Evaluated at index using data within the 180-day period prior to index date. | No | |
| - | Variable indicating any use of insulin using data | Time-dependent | UK: CPRD |
| to insulin | from 180 days prior to index date onwards. ATC codes for insulins in Annex II. | Categorical: | Sweden: SPDR |
| | | Yes | Finland: FPR |
| | Updating from 180 days prior to index date onwards. | No | |
| Metformin | Time updating current exposure status to | Time-dependent | UK: CPRD |
| exposure | metformin based on purchased amounts and daily defined or prescribed dose, using data from 180 days prior to index date onwards. | Categorical: | Sweden: SPDR |
| | | Yes | Finland: FPR |
| | ATC codes for metformin in Annex II. | No | |
| | Updating from 180 days prior to index date onwards. | | |
| | Variable indicating any use of metformin using | Time-dependent | UK: CPRD |
| to metformin | data from 180 days prior to index date onwards. | Categorical: | Sweden: SPDR |
| | ATC codes for metformin in Annex II. | Yes | Finland: FPR |
| | Updating from 180 days prior to index date onwards. | No | |
| Ever exposed | Variable indicating any use of GLP-1 drugs | Time-dependent | UK: CPRD |
| to GLP-1<br>drugs | using data from 180 days prior to index date onwards. | Categorical: | Sweden: SPDR |
| | ATC codes for GLP-1 drugs in Annex II. | Yes | Finland: FPR |
| | Updating from 180 days prior to index date onwards. | No | |

| to | Variable indicating any use of thiazolidinediones using data from 180 days prior to index date onwards. ATC codes for thiazolidinediones in Annex II. Updating from 180 days prior to index date | Time-dependent Categorical: Yes No | UK: CPRD<br>Sweden: SPDR<br>Finland: FPR |
|---|---|---|---|
| to | Variable indicating any use of sulfonylureas using data from 180 days prior to index date | Time-dependent Categorical: | UK: CPRD Sweden: SPDR |
| sulfonylureas | ATC codes for sulfonylureas in Annex II. Updating from 180 days prior to index date onwards. | Yes<br>No | Finland: FPR |
| Ever exposed<br>to other<br>glucose<br>lowering<br>medication | Variable indicating any use of oral glucose lowering drugs other than the study drugs using data from 180 days prior to index date onwards. ATC codes for other glucose lowering drugs in Annex II. Updating from 180 days prior to index date onwards. | Time-dependent<br>Categorical:<br>Yes<br>No | UK: CPRD<br>Sweden: SPDR<br>Finland: FPR |
| Treatment complexity at index | Treatment complexity at index date is categorized by the number of drug classes in concomitant use including study drugs, using data from late80 days prior to index date onwards. Evaluated at index using data from 180 days prior to index date onwards. | Time-fixed Categorical: Monotherapy Dual combination therapy Triple combination therapy or higher | UK: CPRD<br>Sweden: SPDR<br>Finland: FPR |

Table 15 Other non-diabetic concomitant medication use variables

| Variable | Definition | Details | Data source |
|---|---|---|---|
| | Exposure status at index date of any | Time-fixed | UK: CPRD |
| s/diuretics<br>exposure at | antihypertensives/diuretics (including combinations) based on purchased amounts | Categorical: | Sweden: SPDR |
| index date | and daily defined dose using data within 180- | Yes | Finland: FPR |
| | day period prior to index date. | No | |
| | ATC codes for antihypertensives/diuretics in Annex II. | | |
| | Evaluated at index date using data within 180-day period prior to index date. | | |
| Non-steroidal | Exposure status at index date of any NSAID | Time-fixed | UK: CPRD |
| anti-<br>inflammatory | (including combinations) based on purchased amounts and daily defined dose using data | Categorical: | Sweden: SPDR |
| drugs (NSAIDs) | within 180-day period prior to index date. | Yes | Finland: FPR |
| exposure at index date | ATC codes for NSAID in Annex II. | No | |
| macx date | Evaluated at index date using data within 180-day period prior to index date. | | |
| Oral steroids | Exposure status at index date of any oral | Time-fixed | UK: CPRD |
| exposure at index date | steroid (including combinations) based on<br>purchased amounts and daily defined dose<br>using data within 180-day period prior to index<br>date. | Categorical: | Sweden: SPDR |
| macx date | | Yes | Finland: FPR |
| | | No | |
| | ATC codes for oral steroids in Annex II. | | |
| | Evaluated at index date using data within 180-day period prior to index date. | | |
| Statins, fibrates | Exposure status at index date of any statin or | Time-fixed | UK: CPRD |
| exposure at index date | fibrate (including combinations) based on purchased amounts and daily defined dose | Categorical: | Sweden: SPDR |
| mach date | using data within 180-day period prior to | Yes | Finland: FPR |
| | index date. | No | |
| | ATC codes for statins, fibrates in Annex II. | | |
| | Evaluated at index date using data within 180-day period prior to index date. | | |

| companies | | | |
|---|---|---|---|
| Lipid modifying agents exposure at index date | Exposure status at index date of any lipid-modifying agent (including combinations) based on purchased amounts and daily defined dose using data within 180-day period prior to index date. | Time-fixed Categorical: | UK: CPRD<br>Sweden: SPDR |
| | | Yes<br>No | Finland: FPR |
| | ATC codes for lipid modifying agent in Annex II. | | |
| | Evaluated at index date using data within 180-day period prior to index date. | | |
| Zoledronic acid<br>exposure at<br>index date | Exposure status at index date of any zoledronic acid (including combinations) based on purchased amounts and daily defined dose using data within 180-day period prior to index date. | Time-fixed | UK: CPRD |
| | | Categorical: | Sweden: SPDR |
| | | Yes | Finland: FPR |
| | | No | |
| | ATC codes for zoledronic acid in Annex II. | | |
| | Evaluated at index date using data within 180-day period prior to index date. | | |
| Antibiotics | Exposure status at index date of any antibiotic (including combinations) based on purchased amounts, daily defined dose and dose per time estimation using data within 180-day period prior to index date. | Time-fixed | UK: CPRD |
| exposure at index date | | Categorical: | Sweden: SPDR |
| | | Yes | Finland: FPR |
| | | No | |
| | ATC codes for antibiotic in Annex II. | | |
| | Evaluated at index date using data within 180-day period prior to index date. | | |

### 6. PLANNED ANALYSIS

# 6.1. SUMMARY OF STUDY POPULATION IDENTIFICATION

The identification process used to identify the study populations and subgroups will be summarised using population flowcharts including the following information:

- The total number of patients in the source population.
- The number and proportion of patients not meeting inclusion criteria.
- The number and proportion of patients meeting inclusion criteria.
- The number and proportion of patients excluded after applying exclusion criteria.

SEAP for non-interventional study BI Study No: 1245.97

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- The number and proportion of patients included in the study after applying inclusion and exclusion criteria [total study population].
- The number and proportion of patients using empagliflozin (out of total study population) at index date.
- The number and proportion of patients using DPP-4 inhibitors (out of total study population) at index date.

For each of the study countries, a population flowchart similar to Figure 2 will be presented.

#### 6.2. POPULATION DESCRIPTION BEFORE MATCHING

The study population and exposure groups identified in each of the study countries will be described at index date using the following baseline characteristics:

- Demographics and other baseline characteristics at index date Table 11.
- Diabetic complications Table 12 (status at index date).
- Non-diabetic concomitant disease Table 13 (status at index date).
- Diabetic concomitant medication use Table 14 (status at index date).
- Non-diabetic concomitant medication use Table 15 (status at index date).

All continuous variables will be described using standard statistical measures, i.e. range, mean, standard deviation, median, first and third quartile. All categorical variables will be summarized with absolute and relative frequencies.

A summary table will be presented for each of the study countries separately (2 tables). A table template is given in Table 17.

#### 6.3. METHODS ADDRESSING BIAS

Potential biases will be addressed as follows:

- Selection bias and immortal time bias is addressed thru the study design. It include a new user cohort design, a selection of comparator drugs with the same indication and prescribed to patients with potentially similar T2D disease severity, and a definition of exposure and study entry based on information before or at index date.
- Channeling bias is addressed by using propensity score matching to construct balanced exposure groups. In addition, the year of the index date (date of first prescription of the study group) is used as an exact matching criteria.
- Bias due to definitions of exposure, definition of follow-up times and other relevant covariates will be addressed through sensitivity analyses.

• Diagnostic bias will be evaluated and addressed in sensitivity analyses through consideration of the frequency of urine dipstick testing (as captured through albuminuria tests) and stage of cancer at the time of diagnosis (as more early-stage cancers in one group would be suggestive of diagnostic bias).

# 6.4. PROPENSITY SCORE MATCHED COHORTS

#### Matched full cohort

Propensity score matched cohorts will be derived in each country by matching each initiator of empagliflozin at index date with initiators of DPP-4 inhibitors at index date with a variable matching ratio up to 1:3 (1:1 in a sensitivity analysis) using greedy matching methods (cf. Section 6.5). Free or fixed dose combination use of metformin at index date will be used as an exact matching variable.

# Matched metformin-user only cohort

Using the propensity scores computed using the entire cohort, a matched metformin-user only cohort will be derived by matching within a subgroup including only patients using metformin in free or fixed dose combination with the study drugs at index date. Each initiator of empagliflozin at index date will be matched with initiators of DPP-4 inhibitors at index date with a variable matching ratio up to 1:3 using greedy matching methods (cf. Section 6.5).

# 6.5. IMPLEMENTATION OF THE PROPENSITY SCORE MATCHING

# 6.5.1. Estimation of the propensity score

#### **Propensity score model specification**

The propensity score will be estimated using a binary logistic regression model. For all individuals, propensity scores for the comparison empagliflozin vs. DPP-4 inhibitors will be computed at the index date as the probability to receive empagliflozin, conditional on treatment and clinical history up to index date within each stratum.

The resulting propensity score model will be used to create two matched cohorts in each country:

- Matched full cohort, including patients initiating empagliflozin or a DPP-4 inhibitor at index date.
- Matched metformin-user only cohort, including patients using metformin in free or fixed dose combination with empagliflozin or a DPP-4 inhibitor at index date.

#### Variables considered for inclusion in the propensity score model

The following variables will be evaluated at index date and considered for inclusion in the propensity score model:

- Demographics and other baseline characteristics at index date Table 11.
- Diabetic complications Table 12 (status at index date).
- Non-diabetic concomitant disease Table 13 (status at index date).
- Diabetic concomitant medication use Table 14 (status at index date).
- Non-diabetic concomitant medication use Table 15 (status at index date).

# 6.5.2. Matching method

For matching the full cohort, concomitant use of metformin at index date will be an exact matching variable.

Matching will be carried out in several rounds to achieve the highest possible matching ratio given the available data in each country (up to 1:3 matching). In the first round of matching, for each empagliflozin initiator  $i_E$  with index date  $T_{i_E}$ , all individuals initiating DPP-4 inhibitors within 3 months (90 days) before or after  $T_{i_E}$  and with the same status of concomitant metformin use at  $T_{i_E}$  will be eligible as comparators. For UK CPRD data, only individuals from the same database (GOLD or Aurum) as the empagliflozin initiator will be considered as eligible comparators. Of these, the individual with the closest propensity score(s) to that of  $i_E$  within a predefined propensity score interval will be selected (Greedy matching method). In case of ties, the selection will be made randomly. After each round of selection, the selected comparators are then removed from the pool of possible comparators for further selection (sampling without replacement) [5].

The predefined propensity score interval will be calculated based on the standard deviation of the logit of propensity score  $\delta$  multiplied by a coefficient k. The value of the coefficient k will be initially set to 0.2, i.e. using a caliper of 0.2 standard deviations (i.e. 0.2 $\delta$ ). The coefficient k will then be calibrated to ensure at least 99% of empagliflozin initiators have matches from initiators of DPP-4 inihibitors after the first round of propensity score matching [6]. The same calibrated matching caliper  $k\delta$  used in the first matching round will be reused in the second and third matching rounds.

Matching by time-period, based on index dates, enables better control of time-varying confounders including changing prescription patterns for empagliflozin and potential confounding. In case there is a strong time bias in the number of matches per empagliflozin user (e.g., initiators in early years have more matches than initiators from later years), a relaxation of the criteria for matching within time-period will be considered. In addition, the criteria for calibrating coefficient k may be modified if the data does not allow matching of 99% of empagliflozin initiators.

# 6.6. ASSESSING THE QUALITY OF THE MATCHING

# 6.6.1. Propensity score distribution before and after matching and common support region

For each propensity score set (all patient cohort and concomitant metformin users cohort), the propensity score distribution will be plotted for empagliflozin users and DPP-4 inihibitor users before matching (Figure 3). This will be used for visual inspection of the common support region.

The propensity score distribution in non-matched empagliflozin users, matched empagliflozin users, and matched DPP-4 inhibitor users will be plotted for each cohort in each country. Results will be presented in 2 plots similar to Figure 5, one for each of the two propensity score matched cohorts.

# 6.6.2. Assessment of covariate balance before and after matching

The covariates balance between treatment groups before and after matching will be evaluated using:

- Standardized differences (percentage).
- $\chi^2$  test for equality of proportions in dichotomous variables (p-value).
- t-test for equality of means in continuous variables (p-value).

For continuous variables, the standardized difference is defined as

$$d = \frac{(\bar{x}_{empagliflozin} - \bar{x}_{DPP-4 inihibitor})}{\sqrt{\frac{s_{empagliflozin}^2 + s_{DPP-4 inihibitor}^2}{2}} \times 100$$

Where  $\bar{x}_{empagliflozin}$  and  $\bar{x}_{DPP-4\ inihibitor}$  denote the sample mean of the covariate in empagliflozin users at index date and comparison drug users at index date, respectively, while  $s_{empagliflozin}^2$  and  $s_{DPP-4\ inihibitor}^2$  denote the sample variance of the covariate in empagliflozin users at index date and comparison drug users at index date, respectively.

For dichotomous variables, the standardized difference is defined as

$$d = \frac{(\hat{p}_{empagliflozin} - \hat{p}_{DPP-4\ inihibitor})}{\sqrt{\frac{\hat{p}_{empagliflozin}(1 - \hat{p}_{empagliflozin}) + \hat{p}_{DPP-4\ inihibitor}(1 - \hat{p}_{DPP-4\ inihibitor})}}{2}} \times 100$$

Where  $\hat{p}_{empagliflozin}$  and  $\hat{p}_{DPP-4\ inihibitor}$  denote the prevalence of the dichotomous variable in empagliflozin users at index date and DPP-4 inhibitor users at index date, respectively [7]

If a categorical variable is defined with more than two categories (i.e. not dichotomous), each category will be treated as a dichotomous variable when computing the standardized differences.

The balance assessment will be performed with regard to the following covariates:

- Demographics and other baseline characteristics at index date Table 11.
- Diabetic complications Table 12 (status at index date).
- Non-diabetic concomitant disease Table 13 (status at index date).
- Diabetic concomitant medication use Table 14 (status at index date).
- Non-diabetic concomitant medication use Table 15 (status at index date).

Balance in baseline characteristics before and after matching between empagliflozin users at index and the DPP-4 inihibitor users at index will be reported in each country, separately.

All continuous variables will be described using standard statistical measures, i.e. range, mean, standard deviation, median, first and third quartile. All categorical variables will be summarized with absolute and relative frequencies. The standardized differences and p-values for the statistical tests will be also reported.

Results will be reported in 4 tables similar to Table 18.

Standardized difference < 10% will be used as indicator of satisfactory distribution balance after matching [8]. Variables with standardized difference larger than 10% might still exist. The unbalanced variables will be considered as potential confounders and included in the adjustment of Cox's PH model, as described in the comparative analysis (Section 6.7.2). In case a substantial amount of variables remain unbalanced, the PS matching procedure will be re-evaluated by, for example, reducing the caliper width.

## 6.7. AS-TREATED ANALYSIS

#### 6.7.1. Descriptive analysis

Crude incidence rates (IRs) for the outcomes defined in Table 8 will be estimated within each exposure category as defined in Table 5 using Poisson regression.

In addition, stratified IRs will be derived for the following variables:

- Demographics and other baseline characteristics at index date Table 11.

- Diabetic complications Table 12.
- Non-diabetic concomitant disease Table 13.
- Diabetic concomitant medication use Table 14.
- Non-diabetic concomitant medication use Table 15.

Crude IRs will be presented along with 95% CIs. Other descriptive summaries such as number of events and person-time for calculating the IR will be included. Analysis will be performed for each country. Results will be reported as in Table 22.

Kaplan-Meier plots, with 95% CIs, for event-free survival probabilities will be presented for each country for the outcomes defined in Table 8 with exposures as defined in Table 5. Results will be reported as the figure template shown in Figure 6.

Meta-analyses of IRs will be carried out using aggregated data across countries as described in Section 6.7.3.1 and reported as shown in Table 22.

# 6.7.2. Comparative analysis

Hazard ratios (HRs) for the outcomes defined in Table 8 will be estimated for PS matched cohorts using Cox's PH model with time-varying covariates, if model pre-requisites are fulfilled. HRs will be presented along with 95% CIs. Proportional hazards assumptions for time-fixed exposure variables will be assessed for each model by plotting scaled Schoenfeld residuals.

The comparative analyses will be performed separately for the matched full cohort and matched metformin-user cohort.

#### Crude model

Crude HRs are calculated using a Cox PH model with as-treated exposure (as defined in Section 5.1.7) as the only included variable.

HRs estimated using the crude model will be presented along with 95% CIs. A table template for the result is given in Table 23. Analysis will be performed separately for each country.

Crude HRs with 95% CIs will be collected from all study countries to carry out metaanalyses as described in Section 6.7.3.2. Results will be reported as in Figure 8.

#### Base model

Based on the crude model, the base model will be further adjusted with the unbalanced covariates at index date (standard difference  $\geq 10\%$ ) among the variables included in the propensity score model (Section 6.6). The inclusion of adjusting variables will be considered based on data availablity as described in Section 10.

HRs estimated using the base model will be presented along with 95% CIs. A table template for the result is given in Table 24. Analysis will be performed separately for each country. HRs with 95% CIs estimated using base model will be collected from all study countries to carry out meta-analyses as described in Section 6.7.3.2. Results will be reported as in Figure 8.

### **Adjusted model**

The base model will be further adjusted with selected time-dependent variables. The following time-dependent variables will be initially considered for inclusion (as detailed in Section 9) in the adjusted Cox's PH model:

- HbA1c value (as defined in Table 11)
- Kidney or genitourinary stones (as defined in Table 13)
- UTI or pyelonephritis (as defined in Table 13)
- Ever exposed to insulin (as defined in Table 14)
- Ever exposed to metformin (as defined in Table 14)

- Ever exposed to other glucose lowering medication (as defined in Table 14)
- Ever exposed to GLP-1 drugs (as defined in Table 14)
- Ever exposed to thiazolidinediones (as defined in Table 14)
- Ever exposed to sulfonylureas (as defined in Table 14)

HRs estimated using the adjusted model with time-dependent covariates will be presented along with 95% CIs. A table template for the result is given in Table 25. Analysis will be performed and model adjustment will be applied separately for each country.

Adjusted HRs with 95% CIs will be collected from all study countries to carry out metaanalyses as described in Section 6.7.3.2. Results will be reported as in Figure 8.

### Handling of model convergence failure

For outcomes with a small number of events, converge failure of multivariable Cox PH regression model may happen if there are no events for a particular combination of covariate values. Thus, a minimum of 5 outcome events per category of a variable is required for it to be included in the Cox model. In case of persisting model convergence failure while meeting this minimum requirement, the included covariates will be removed sequentially based on the rank of their PS standardised differences. The covariate with the smallest standardised difference will be removed iteratively until the model converges. In case of ties in selection, the choice is made randomly. The removed covariates will be reported along with the HR estimates.

#### 6.7.3. META-ANALYSES

Meta-analyses will be carried out when there is no relevant heterogeneity of variable definitions and effect size of outcomes with respect to primary exposures among country-specific analyses. Country-level effect-sizes will be pooled using meta-analysis models to compute pooled effect-size estimates.

#### 6.7.3.1. META-ANALYSIS OF DESCRIPTIVE ANALYSES

#### **Pooled incidence rates**

For each outcome, the aggregated number of events and person-time at risk will be collected from all study countries to estimate the pooled IRs and their 95% CIs.

The pooled IRs for all K countries will be estimated as

$$IR_{pooled} = \frac{\sum_{k=1}^{K} x_k}{\sum_{k=1}^{K} t_k}$$

where  $x_k$  and  $t_k$  are the number of events and the person-time at risk in each country k. 95% CIs will be estimated using Poisson regression and reported similarly using Table 22.

#### 6.7.3.2. META-ANALYSIS OF COMPARATIVE ANALYSIS

Meta-analyses will combine the estimates of adjusted HRs across countries using the inverse-variance method. Log-transformed HRs and their standard errors will be collected to calculate pooled HR estimates using random-effects models. Pooled HRs and their 95% CI will be reported using forest plots. In a sensitivity analysis, pooled HRs will be estimated using fixed-effect models.

## **Between-study heterogeneity**

Prior to conducting meta-analyses, heterogeneity across the countries in terms of study design and conduct will be assessed. Specifically, the variability in population characteristics (including data availability), in pre- and post- PS matching balance in baseline characteristics between cohorts, as well as in observed incidence rates will be examined. If needed, changes in study population selection criteria or other analysis parameters will be considered to reduce such heterogeneity.

Statistical heterogeneity between country-level estimates will be estimated using Higgins' and Thompson's  $I^2$  [9] and the moment-based estimate of  $\tau^2$ .

Both  $I^2$  and  $\tau^2$  are derived using Cochran's Q statistic defined as

$$Q = \sum_{k=1}^{K} w_k \left( \hat{\theta}_k - \frac{\sum_{k=1}^{K} w_k \hat{\theta}_k}{\sum_{k=1}^{K} w_k} \right)^2; w_k = \frac{1}{s_k^2}$$

where  $\hat{\theta}_k$  denotes the log-transformed per-country HR estimate,  $s_k^2$  its variance,  $w_k$  the corresponding weight from the country-level study k calculated as the inverse of variance  $s_k^2$ .

# $I^2$ statistic

 $I^2$  is the percentage of variability in the treatment estimates which is attributable to heterogeneity between studies rather than to sampling error.  $I^2$  is formulated as

$$I^2 = max \left\{ 0, 1 - \frac{K-1}{Q} \right\}$$

where *Q* is Cochran's Q statistic and *K* is the number of the per-country studies.

 $I^2$  and its 95% CIs are used to assess the importance of between study heterogeneity as follows:

- 0% to 40%: might not be important
- 30% to 60%: may represent moderate heterogeneity
- 50% to 90%: may represent substantial heterogeneity
- 75% to 100%: considerable heterogeneity

SEAP for non-interventional study BI Study No: 1245.97

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

 $I^2$  is sensitive to the precision of the included studies, with higher  $I^2$  associated with increased precision in individual studies.

## $\tau^2$ statistic

The  $\tau^2$  statistic represents the variance of the distribution of the true effect-sizes.  $\tau^2$  will be calculated using the DerSimonian and Laird estimate:

$$\hat{\tau}^2 = max \left\{ 0, \frac{Q - (K - 1)}{\sum_{k=1}^{K} w_k - \frac{\sum_{k=1}^{K} w_k^2}{\sum_{k=1}^{K} w_k}} \right\}; w_k = \frac{1}{s_k^2}$$

where  $w_k$  denotes the corresponding weight from the per-country study k, and  $s_k^2$  is the variance of HR estimate of per-country study k.

 $\tau^2$  is insensitive to the number of studies or to their precision but can be difficult to interpret. It is however expressed at the same scale as square of the effect size; hence its 95% CI represents the estimated range of true effect sizes.

#### Random-effects model

The random-effects model considers the observed per-country effect sizes as randomly sampled from a distribution of true effect sizes. The pooled effect size estimated by the model represents the mean of this distribution of true effect sizes.

In addition to the sampling error (squared as variance  $s_k^2$ ), the random-effects model takes into account the variance of the distribution of the true effects, which is estimated as between-study heterogeneity tau-squared  $\tau^2$ . The weight  $w_k$  for each country k is calculated with  $\tau^2$  as an additional scaling factor, resulting in the adjusted random-effects weights  $w_k^*$ .

$$w_k^* = \frac{1}{s_k^2 + \tau^2}$$

The pooled HR estimate  $\hat{\theta}$  is calculated using adjusted weights  $w_k^*$ .

$$\hat{\theta} = \frac{\sum_{k=1}^{K} \hat{\theta}_k w_k^*}{\sum_{k=1}^{K} w_k^*}$$

For each meta-analysis, pooled and country-level results will be presented in forest plots similar to Figure 8 showing the following items:

- Country identifier
- Number of events (IR/1000 person years) per study group
- HR and 95% CI for each country (on log scale)
- The weight (%) assigned to each country
- The estimated pooled HR and its 95% CI using a random-effect models (on log scale)

- Total number of patients per study group
- Average follow-up time in person years
- Between-study heterogeneity  $\tau^2$  and its 95% CI
- The  $I^2$  statistics and its 95% CI







SEAP for non-interventional study BI Study No: 1245.97

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6.10. LIST OF PLANNED ANALYSIS

Table 16 List of planned analyses.

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Population identification | | | | |
| Summary of the process used to identify the study | Country specific analysis | N/A | N/A | Figure 2 |
| populations and study treatment groups. | (3 figures, one for each country) | 1 1/1 1 | | |
| Population description b | efore matching | | | |
| Description of patient baseline characteristics | Country specific analysis | | N/A | Table 17 |
| for the study population<br>and the study treatment<br>groups before matching. | (3 tables, one for each country) | N/A | | |
| Assessment of covariate | balance before matching | | | |
| Balance assessment for baseline characteristics between empagliflozin | Country specific analysis | N/A | N/A | Table 18 |
| users at index and DPP-4 inhibitors users at index before matching. | (3 tables, one for each country) | | | |
| | pensity score distribution | | | |
| Propensity score distribution plot for | Country specific analysis | | N/A | Figure 3 |
| empagliflozin users at index and DPP-4 inhibitors users at index. | (3 figures, one for each country) | N/A | | |
| Assessing the quality of t | he matching | | | |
| Balance assessment for baseline characteristics between empagliflozin | Country specific analysis | NI/A | N/A | Table 18 |
| users at index and DPP-4 inhibitors users at index after matching. | (3 tables, one for each country) | N/A | 11/12 | Table 18 |
| Standardized differences plot before and after PS matching for | Country specific analysis | N/A | N/A | Figure 4 |
| empagliflozin users at index vs. DPP-4 inhibitors users at index | (3 figures, one for each country) | IN/A | 1V/A | riguit 4 |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Propensity score distribution in non-matched empagliflozin users at index date matched empagliflozin users at index and matched DPP-4 inhibitors users at index. | Country specific analysis (3 figures, one for each country) | N/A | N/A | Figure 5 |
| Propensity score assessment distribution | Country specific analysis (3 tables, one for each country) | N/A | N/A | Table 19 |
| Primary objectives:<br>Descriptive analysis | | | | |
| Stratified incidence rates | Using matched cohorts Country specific analysis (9 tables, 3 outcomes x 3 countries) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 22 |
| Meta-analysis of incidence rates | Using pooled number of outcome events and persontime from all study countries (3 tables, 3 outcomes) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 22 |
| Kaplan-Meier survival probability plots | Using matched cohorts Country specific analysis (9 figures, 3 outcomes x 3 countries) | As treated exposure definition | Main outcomes-<br>Table 8 | Figure 6 |
| Primary objectives:<br>Comparative analysis | | | | |
| Hazard ratio estimates using crude model | Using matched cohorts Country specific analysis (18 tables, 2 cohorts x 3 outcomes x 3 countries | As treated exposure definition | Main outcomes-<br>Table 8 | Table 23 |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Meta-analysis of crude<br>HR estimates | Using adjusted HR estimates and 95% CIs from all study countries | As treated exposure definition | Main outcomes-<br>Table 8 | Figure 8 |
| | (2 cohorts: 6 figures, 3 outcomes) | | | |
| Hazard ratio estimates using the base model | Using matched cohorts<br>Country specific analysis | As treated exposure definition | Main outcomes-<br>Table 8 | Table 23 |
| | (18 tables, 2 cohorts x 3 outcomes x 3 countries) | | | |
| Meta-analysis of HR estimates using the base model | Using adjusted HR estimates and 95% CIs from all study countries | As treated exposure definition | Main outcomes-<br>Table 8 | Figure 8 |
| | (2 cohorts: 6 figures, 3 outcomes) | | | |
| Hazard ratio estimates using the adjusted model | Using matched cohorts Country specific analysis | As treated exposure definition | Main outcomes-<br>Table 8 | Table 25 |
| | (18 tables, 2 cohorts x 3 outcomes x 3 countries) | | | 14010 20 |
| Meta-analysis of adjusted HR estimates | Using adjusted HR estimates and 95% CIs from all study countries | As treated exposure definition | Main outcomes-<br>Table 8 | Figure 8 |
| | (2 cohorts: 6 figures, 3 | | | |
| Stratified analysis | outcomes) | | | |
| Straulieu alialysis | Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Stratified by treatment complexity at index. | As treated exposure definition | Main outcomes-<br>Table 8 | T 11 25 |
| | (27 tables, 3 outcomes x 3 strata by treatment complexity at index x 3 countries) | | | Table 25 |

SEAP for non-interventional study BI Study No: 1245.97

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| | Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Stratified by PS quartiles at index. | As treated exposure definition | Main outcomes-<br>Table 8 | Table 25 |
| | (36 tables, 3 outcomes x 4 strata by propensity score quartiles x 3 countries) | | | |
| | Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Stratified by age category at index. | As treated exposure | Main outcomes-<br>Table 8 | Table 25 |
| | (63 tables, 3 outcomes x 7 strata by age category x 3 countries) | definition | | |
| | Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Stratified by gender. | As treated exposure | Main outcomes-<br>Table 8 | Table 25 |
| | (18 tables, 3 outcomes x 2 strata by gender x 3 countries) | definition | | |
| | Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Stratified by insulin use at index. | As treated exposure | Main outcomes-<br>Table 8 | Table 25 |
| | (18 tables, 3 outcomes x 2 strata by insulin use at index x 3 countries) | definition | | |
| Meta-analyses for adjusted HR estimates | Using adjusted HR estimates and 95% CIs from all study countries. | | | |
| | For each stratification variable listed above. | As treated exposure definition | Main outcomes-<br>Table 8 | Figure 8 |
| | (54 figures, 3 outcomes x (3+4+7+2+2) strata) | | | |
| Secondary objectives:<br>Descriptive analysis | | | | |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Stratified incidence rates | Using matched cohorts Country specific analysis (9 tables, 3 outcomes x 3 countries) | Cumulative<br>exposure<br>dose of<br>empaglifloz<br>in | Main outcomes-<br>Table 8 | Table 30 |
| Stratified incidence rates | Using empagliflozin users subgroup Country specific analysis (9 tables, 3 outcomes x 3 countries) | Empaglifloz<br>in daily<br>dose | Main outcomes-<br>Table 8 | Table 31 |
| Stratified incidence rates | Using empagliflozin users subgroup Country specific analysis (9 tables, 3 outcomes x 3 countries) | Cumulative exposure duration to empaglifloz in | Main outcomes-<br>Table 8 | Table 32 |
| Meta-analysis of incidence rates | Using pooled number of outcome events and persontime from all study countries (9 tables, 3 outcomes x 3 secondary exposure definitions) | The secondary exposure definitions listed above | Main outcomes-<br>Table 8 | Table 30-<br>Table 32 |
| Secondary objectives:<br>Comparative analysis | , | | | |
| Hazard ratio estimates using adjusted model | Using matched cohorts Country specific analysis (9 tables, 3 outcomes x 3 | Cumulative exposure dose of empaglifloz in | Main outcomes-<br>Table 8 | Table 26 |
| | Countries) Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Country specific analysis (9 tables, 3 outcomes x 3 countries) | Empaglifloz<br>in daily<br>dose | Main outcomes-<br>Table 8 | Table 27 |
| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| | Using matched cohorts | Cumulative | | |
| Hazard ratio estimates using adjusted model | Country specific analysis | exposure duration to | Main outcomes-<br>Table 8 | Table 28 |
| using adjusted model | (9 tables, 3 outcomes x 3 countries) | empaglifloz<br>in | | |
| Meta-analysis of adjusted | Using adjusted HR estimates with 95% CIs from all study countries | 3 secondary exposure | Main outcomes- | |
| HR estimates | (9 figures, 3 outcomes x 3 secondary exposure | definitions<br>listed above | Table 8 | Figure 8 |
| Sensitivity analysis:<br>NCC study design | | | | |
| Balance assessment for baseline characteristics between matched cases and controls. | Country specific analysis (3 tables, one for each country) | N/A | N/A | Table 33 |
| Odds ratio using | Nested case-control study design. | As treated | All cancer cases | |
| conditional logistic regression | (3 tables, 1 outcome (all cancer cases) x 3 countries) | exposure<br>definition | defined in Table 8 | Table 34 |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Sensitivity analysis:<br>Adjusting for time-depen | dent confounding | | | |
| | Using matched cohorts | | | |
| Hazard ratio estimates using marginal structural model | MSM using IPTW. | As treated exposure definition | Urinary tract cancer as defined in Table | Table 35 |
| | (3 tables, 1 outcome x 3 countries) | | 8 | |
| Meta-analysis of adjusted<br>HR estimates using<br>MSM | Using adjusted HR estimates with 95% CIs from all study countries | As treated exposure definition | Urinary tract cancer as defined in Table 8 | Figure 8 |
| | (1 figure, 1 outcome) | | | |
| Sensitivity analysis:<br>Exposures | | | | |
| Hazard ratio estimates | Using matched cohorts | Intention to treat | Urinary tract cancer as | T 11 25 |
| using adjusted model | (3 tables, 1 outcome x 3 countries) | exposure definition | defined in Table<br>8 | Table 25 |
| Meta-analysis of adjusted | Using adjusted HR estimates with 95% CIs from all study countries | Intention to treat | Urinary tract cancer as | Figure 8 |
| HR estimates | (1 figure, 1 outcome) | exposure<br>definition | defined in Table<br>8 | riguic o |
| Sensitivity analysis:<br>Grace period | | | | |
| | Using matched cohorts | | | |
| Hazard ratio estimates using adjusted model | Allowed gaps between exposure episodes extended to 90 days | Intention to treat exposure definition | Urinary tract<br>cancer as<br>defined in Table<br>8 | Table 25 |
| | (3 tables, 1 outcome x 3 countries) | <del></del> | | |
| | Using adjusted HR estimates with 95% CIs from all study | Intention to | Urinary tract | |
| Meta-analysis of adjusted HR estimates | countries | treat | Urinary tract cancer as defined in Table | Figure 8 |
| TIX estimates | (1 figure, 1 outcome) | exposure<br>definition | 8 | |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Sensitivity analysis:<br>Outcomes | | | | |
| Crude incidence rates | Using matched cohorts Country specific analysis (9 tables, 3 outcomes x 3 countries) | As treated exposure definition | Further outcomes-Table 9 | Table 29 |
| Hazard ratio estimates using adjusted model | Using matched cohorts (3 tables, 3 outcomes) | As treated exposure definition | Further outcomes-Table 9 | Table 25 |
| TNM staging at diagnosis | Using matched cohorts (9 tables, 3 outcomes x 3 countries) | As treated exposure definition | Further outcomes-Table 10 | Table 21 |
| Albuminaria tests each year | Using matched cohorts (3 tables, 3 countries) | As treated exposure definition | NA | Table 36 |
| Sensitivity analysis:<br>Extended latency period | , | | | |
| Hazard ratio estimates using adjusted model | Using matched cohorts Duration of latency period is extended to 12 months. (3 tables, 1 outcome x 3 countries) | As treated exposure definition | Urinary tract<br>cancer as<br>defined in Table<br>8 | Table 25 |
| Meta-analysis of adjusted HR estimates | Using adjusted HR estimates with 95% CIs from all study countries (1 figure, 1 outcome) | As treated exposure definition | Urinary tract cancer as defined in Table 8 | Figure 8 |
| Hazard ratio estimates using adjusted model | Using matched cohorts Discontinuation is 6 months after last day of medication or switch. (3 tables, 1 outcome x 3 countries) | As treated exposure definition | Urinary tract<br>cancer as<br>defined in Table<br>8 | Table 25 |
| Meta-analysis of adjusted HR estimates (discontinuation is 6 months after last day of medication or switch) | Using adjusted HR estimates with 95% CIs from all study countries (1 figure, 1 outcome) | As treated exposure definition | Urinary tract cancer as defined in Table 8 | Figure 8 |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Sensitivity analysis: Inclusion of the Aurum ( | CPRD database | | | |
| Description of patient<br>baseline characteristics<br>for the UK, stratified by<br>CPRD database | CPRD specific analysis (1 table) | N/A | N/A | Table 37 |
| Stratified incidence rates | Using UK matched cohorts (3 tables, 3 outcomes x 1 country) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 38 |
| Hazard ratio estimates<br>using crude model after<br>adding CPRD database<br>as a stratification variable | Using UK matched cohorts (3 tables, 3 outcomes x 1 country) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 39 |
| Hazard ratio estimates using the base model after adding CPRD database as a stratification variable | Using matched cohorts Only for the UK (3 tables, 3 outcomes x 1 table) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 40 |
| Hazard ratio estimates using the adjusted model after adding CPRD database as a stratification variable | Using matched cohorts Only for the UK (3 tables, 3 outcomes x 1 table) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 41 |
| Hazard ratio estimates using the crude model, stratified by UK-CPRD databases | Using UK matched cohorts (3 tables, 3 outcomes x 1 country) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 42 |
| Hazard ratio estimates using the base model, stratified by UK-CPRD databases | Using UK matched cohorts (3 tables, 3 outcomes x 1 country) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 43 |
| Hazard ratio estimates using the base model, stratified by UK-CPRD databases | Using UK matched cohorts (3 tables, 3 outcomes x 1 country) | As treated exposure definition | Main outcomes-<br>Table 8 | Table 44 |
| Sensitivity analysis:<br>Meta-analysis using fixed | • | | | |

| Analysis | Details | Exposure definition | Outcomes | Template |
|---|---|---|---|---|
| Meta-analysis of adjusted HR estimates using a fixed-effect model | Using adjusted HR estimates and 95% CIs from all study countries | As treated exposure definition | Main outcomes-<br>Table 8 | Figure 9 |
| | (3 figures, 3 outcomes) | | | |

#### 7. DATA MANAGEMENT

will collect electronic patient records and comply with procedures that include checking electronic files, maintaining security and data confidentiality, following analyses plans, and performing quality checks for all programs.

will maintain any patient-identifying information securely on site according to up-to-date standard operating procedures.

will also maintain appropriate data storage, and archiving procedures will be

#### 8. STATISTICAL SOFTWARE

followed with periodic backup of files.

R language (http://www.r-project.org) will be used in statistical analysis for creating tabulations and graphics as well as in all statistical modelling. R language is described in more details in report "R: Regulatory Compliance and Validation Issues: A Guidance Document for the Use of R in Regulated Clinical Trial Environments" (www.r-project.org/doc/R-FDA.pdf, read 21 December 2016)[12].

#### 9. MISSING DATA

A high frequency of missing values is not expected for most variables, with the possible exception of lifestyle and biological measurement variables. For the medical history conditions / comorbidities to be collected for inclusion in the propensity score, the absence of a code for a condition will be interpreted as an absence of the event.

If a variable is missing for only some of the patients, a missing data category will be added and utilized in the analysis. If a variable is missing for more than 50% of patients, removal of the variable from the relevant model or analysis (propensity score, multivariable Cox's regression, NCC matching) will be considered.

#### 10. QUALITY CONTROL

The data analysis will be conducted as specified in the SEAP. The principal investigator, the co-investigators and the sponsors of the study must approve all revisions to the SEAP. All major changes to the SEAP shall be properly documented as SEAP amendments and when necessary such SEAP amendments will be implemented in the study protocol and delivered to relevant ethics committees and register holders.

will be the registered holder for the retrieved Swedish, Finnish and UK data, also with the responsibility for destroying the data after the study, when legally possible. A quality control will be performed on the retrieved register data, including the inclusion of compulsory variables, such as SID and main diagnosis, in the delivered register data. If data are missing or incorrect, the dataset is sent back to the register holder for correction.

All processes from data management leading to dissemination of study results will undergo quality control checks for programs, result tables and written text, according to standard Operating Procedures and project-specific instructions RWI\_WI\_EPI0010 "Non-Interventional Study and Low Intervention Clinical Trial Report Development", RW\_PI\_OP-401.01\_003\_01 "Programming and statistical analysis", and RW\_PI\_OP-406.01\_003\_01 "Programming validation". A detailed audit trail of all documents (programs, result tables, reports) along with quality control processes will be maintained.

All programs for data management and data analyses written by study statistician(s) will be self-documenting with comments about the data handling process, the population selection and the analysis performed by the program. The documentation will be sufficient for another statistician to be able to repeat the program. A statistician other than the one who writes the program will carry out quality control checks of these programs. The programming QC will be performed for all programs related to the database, its individual datasets from different registers and statistical analyses. The QC will be documented with the following information:

- Name of the program
- Purpose of the program
- Name of the programmer
- Validation status and date of validation
- Updates and dates of updates
- Name of the QC statistician
- QC findings or comments
- Date of QC

The statistician responsible for the QC of a program will ensure that:

- The correct dataset and population has been used
- The analysis is carried out according to the SEAP
- The analysis results are consistent
- The output is in line with the table shells in the SEAP
- The analysis can be interpreted in both statistical and clinical terms.

All QC findings by the QC statistician will be documented, and corrections are made to the programs accordingly. All changes are documented as updates to the original program.

The raw dataset and statistical programs used for generating the data included in the final study report will be kept in electronic format and be available for auditing and inspection.

As the register holder of the study register is in charge of archiving and deleting the data. Secure archives will be maintained for the orderly storage and retrieval of all study related material. An index shall be prepared to identify the archived contents and their location. Access to the archives will be controlled and limited to authorised personnel only. Access to the study data cannot be given to any third parties, neither the study data can be used to other purposes than prescribed in the study protocol. All requests to use the study data for other purposes than mentioned in the study protocol must be subjected to appropriate data permit processes.

### 11. REFERENCES

- [1] S. Schneeweiss, "A basic study design for expedited safety signal evaluation based on electronic healthcare data," *Pharmacoepidemiol Drug Saf*, vol. 19, no. 8, pp. 858–868, Aug. 2010, doi: 10.1002/pds.1926.
- [2] E. Patorno *et al.*, "Observational studies of the association between glucose-lowering medications and cardiovascular outcomes: addressing methodological limitations," *Diabetologia*, vol. 57, no. 11, pp. 2237–2250, Nov. 2014, doi: 10.1007/s00125-014-3364-z.
- [3] CPRD, "Clinical Practice Research Datalink," 2021. https://www.cprd.com/ (accessed Nov. 04, 2021).
- [4] L. Pazzagli *et al.*, "Methods for constructing treatment episodes and impact on exposure-outcome associations," *Eur J Clin Pharmacol*, vol. 76, no. 2, pp. 267–275, Feb. 2020, doi: 10.1007/s00228-019-02780-4.
- [5] J. A. Rassen, A. A. Shelat, J. Myers, R. J. Glynn, K. J. Rothman, and S. Schneeweiss, "One-to-many propensity score matching in cohort studies," *Pharmacoepidemiol Drug Saf*, vol. 21 Suppl 2, pp. 69–80, May 2012, doi: 10.1002/pds.3263.
- [6] P. C. Austin, "Optimal caliper widths for propensity-score matching when estimating differences in means and differences in proportions in observational studies," *Pharm Stat*, vol. 10, no. 2, pp. 150–161, Apr. 2011, doi: 10.1002/pst.433.
- [7] P. C. Austin, "Balance diagnostics for comparing the distribution of baseline covariates between treatment groups in propensity-score matched samples," *Statistics in Medicine*, vol. 28, no. 25, pp. 3083–3107, 2009, doi: 10.1002/sim.3697.
- [8] S.-L. T. Normand *et al.*, "Validating recommendations for coronary angiography following acute myocardial infarction in the elderly: A matched analysis using propensity scores," *Journal of Clinical Epidemiology*, vol. 54, no. 4, pp. 387–398, Apr. 2001, doi: 10.1016/S0895-4356(00)00321-8.
- [9] J. P. T. Higgins and S. G. Thompson, "Quantifying heterogeneity in a meta-analysis," *Statistics in Medicine*, vol. 21, no. 11, pp. 1539–1558, Jun. 2002, doi: 10.1002/sim.1186.
- [10] V. Essebag, R. W. Platt, M. Abrahamowicz, and L. Pilote, "Comparison of nested case-control and survival analysis methodologies for analysis of time-dependent exposure," *BMC Medical Research Methodology*, vol. 5, no. 1, p. 5, Jan. 2005, doi: 10.1186/1471-2288-5-5.
- [11] S. R. Cole and M. A. Hernán, "Constructing Inverse Probability Weights for Marginal Structural Models," *Am J Epidemiol*, vol. 168, no. 6, pp. 656–664, Sep. 2008, doi: 10.1093/aje/kwn164.
- [12] "R: Regulatory Compliance and Validation Issues: A Guidance Document for the Use of R in Regulated Clinical Trial Environments." www.r-project.org/doc/R-FDA.pdf

## Annex I

# Diagnosis and operation codes.

The list of diagnosis and operation codes will be provided in separate documents.

• Annex 1.1 - Diagnosis and operation codes for CPRD Gold



Annex 1.1.zip

Annex 1.2 - Diagnosis and operation codes for CPRD Aurum



Annex 1.2.zip

• Annex 1.3 - Diagnosis and operation codes for Finland and Sweden



Annex 1.3.xlsx

## Boehringer Ingelheim SEAP for non-interventional study BI Study No: 1245.97


### **Annex II**

## **ATC** codes used to define treatments

The corresponding READ codes used to define treatments for CPRD will be provided in a separate document.

Annex 2.1 - READ codes for treatment definition for CPRD Gold



Annex 2.2 - READ codes for treatment definition for CPRD Aurum



Annex 2.2.zip

| Drug Group | ATC codes |
|---|---|
| Empagliflozin alone or in combination with | |
| metformin; excluding fixed dose combinations with | |
| drugs other than empagliflozin | |
| Empagliflozin | A10BK03 (previously A10BX12) |
| metformin and empagliflozin | A10BD20 |
| Other SGLT-2 inhibitors; excluding empagliflozin | |
| and excluding fixed-dose combinations with DPP-4 | |
| inhibitors | |
| Dapagliflozin | A10BK01 (previously: A10BX09) |
| Canagliflozin | A10BK02 (previously: A10BX11) |
| Ertugliflozin | A10BK04 |
| Ipragliflozin | A10BK05 |
| metformin and dapagliflozin | A10BD15 |
| metformin and canagliflozin | A10BD16 |
| Metformin and ertugliflozin | A10BD23 |
| DPP-4 inhibitors; excluding fixed-dose combinations | |
| with SGLT-2 inhibitors | |
| Sitagliptin | A10BH01 |
| Vildagliptin | A10BH02 |
| Saxagliptin | A10BH03 |
| Alogliptin | A10BH04 |
| Linagliptin | A10BH05 |
| Evogliptin | A10BH07 |
| Gemigliptin | A10BH06 |
| sitagliptin and simvastatin | A10BH51 |
| gemigliptin and rosuvastatin | A10BH52 |
| metformin and sitagliptin | A10BD07 |
| metformin and vildagliptin | A10BD08 |
| pioglitazone and alogliptin | A10BD09 |
| metformin and saxagliptin | A10BD10 |
| metformin and linagliptin | A10BD11 |
| pioglitazone and sitagliptin | A10BD12 |
| metformin and alogliptin | A10BD13 |
| metformin and gemigliptin | A10BD18 |
| metformin and evogliptin | A10BD22 |
| Fixed dose combinations of SGLT-2 inhibitors with | |
| DPP-4 inhibitors | |
| linagliptin and empagliflozin | A10BD19 |
| saxagliptin and dapagliflozin | A10BD21 |
| Sitagliptin and ertugliflozin | A10BD24 |
| metformin, saxagliptin and dapagliflozin | A10BD25 |
| Insulin | |
| Insulins and analogues | A10A |
| Metformin (alone or in fixed dose combinations) | |
| Metformin | A10BA02 |
| metformin and sulfonylureas | A10BD02 |
| metformin and rosiglitazone | A10BD03 |
| metformin and pioglitazone | A10BD05 |
| metformin and sitagliptin | A10BD07 |
| metformin and vildagliptin | A10BD08 |

| | 110DD10 |
|----------------------------------------------------|-----------|
| metformin and saxagliptin | A10BD10 |
| metformin and linagliptin | A10BD11 |
| metformin and alogliptin | A10BD13 |
| metformin and repaglinide | A10BD14 |
| metformin and dapagliflozin | A10BD15 |
| metformin and canagliflozin | A10BD16 |
| metformin and acarbose | A10BD17 |
| metformin and gemigliptin | A10BD18 |
| metformin and empagliflozin | A10BD20 |
| metformin and evogliptin | A10BD22 |
| metformin and ertugliflozin | A10BD23 |
| metformin, saxagliptin and dapagliflozin | A10BD25 |
| Other glucose lowering medication | |
| exenatide | A10BX04 |
| liraglutide | A10BX07 |
| lixisenatide | A10BX10 |
| albiglutide | A10BX13 |
| repaglinide | A10BX02 |
| nateglinide | A10BX03 |
| mitiglinide | A10BX08 |
| metformin and repaglinide | A10BD14 |
| pramlintide | A10BX05 |
| benfluorex | A10BX06 |
| guar gum | A10BX01 |
| GLP-1 drugs | ATODAOT |
| Glucagon-like peptide-1 receptor (GLP-1) analogues | A10BJ |
| Thiazolidinediones | Alobi |
| Thiazolidinediones | A10BG |
| glimepiride and rosiglitazone | A10BD04 |
| metformin and rosiglitazone | A10BD03 |
| $\mathcal{E}$ | |
| glimepiride and pioglitazone | A10BD06 |
| metformin and pioglitazone | A10BD05 |
| pioglitazone and alogliptin | A10BD09 |
| pioglitazone and sitagliptin | A10BD12 |
| Sulfonylureas | |
| Sulfonylureas | A10BB |
| phenformin and sulfonylreas | A10BD01 |
| metformin and sulfonylreas | A10BD02 |
| glimepiride and rosiglitazone | A10BD04 |
| glimepiride and pioglitazone | A10BD06 |
| glymidine | A10BC01 |
| tolbutamide | V04CA01 |
| Antihypertensives/diuretics | |
| Antihypertensives | C02 |
| Diuretics | C03 |
| Beta blocking agents | C07 |
| Calcium channel blockers | C08 |
| Agents acting on the renin-angiotensin system | C09 |
| minoxidil | D11AX01 |
| clonidine | N02CX02 |
| clonidine | S01EA04 |
| violitatiiv | ~VIL/10 I |

| - |
|---------------------------------------|
| · |

# **Annex III**

# Tables and figures templates

Figure 2 Flowchart of the study population and study subgroups identification in [Study country].



Abbreviations: DPP-4, dipeptidyl peptidase-4; T2DM, Type 2 diabetes mellitus.

**Definitions:** Index date, the date of first purchase/prescription of empagliflozin or DPP-4 between August 1, 2014 and June 30, 2020.

Table 17 Patients baseline characteristics in each of the study groups and in the total study population in [Study country].

| | , , , | | |
|---|---|---|---|
| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study population |
| | N | N | (Total) |
| Age at index (years) | | | |
| 18-49 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 50-64 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 65-69 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 70-74 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 75-79 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 80-84 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 85 and over | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Sex | | | |
| Male | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Female | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Highest level of education | | | |
| Compulsory | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Upper secondary | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Post secondary | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Disposable income, Individual | | | |
| < Q1 | N (x.xx%) | N (x.xx%) | N (x.xx%) |


| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| Q1 – Q2 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q2 – Q3 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq Q3$ | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Disposable income, family | | | |
| < Q1 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q1 – Q2 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q2 – Q3 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥ Q3 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Marital status | | | |
| Registered partnership (incl. married) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Widowed | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Separated | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Single | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Calendar year of index date | | | |
| 2014 | N(x.xx%) | N (x.xx%) | N (x.xx%) |
| 2015 | N(x.xx%) | N (x.xx%) | N (x.xx%) |
| 2016 | N(x.xx%) | N (x.xx%) | N (x.xx%) |

| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| 2017 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2018 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2019 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2020 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2021 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Duration of look-back period | | | |
| 1 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2-5 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 6-9 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 10 and over | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Time since first diabetes diagnosis at index date | | | |
| <q1< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td></q1<> | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq$ (x <q2< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td></q2<> | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq$ (x <q3< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td></q3<> | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥( | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |

| | | 1 | |
|---|---|---|---|
| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
| | N | N | (Total) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Duration of treated diabetes at index | | | |
| date | | | |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Diabetes treatment complexity at index | | | |
| date | | | |
| Monotherapy | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Dual combination therapy | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Triple combination therapy | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Insulin use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Insulin use at index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Metformin use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Metformin use at index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |


| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Oral glucose lowering drugs use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Oral glucose lowering drugs use at index | | | |
| date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Sulfonylureas use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Sulfonylureas use at index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Thiazolidinediones use prior to index | | | |
| date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Thiazolidinediones use at index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |

| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| GLP-1 use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| GLP-1 use at index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic complications prior | | | |
| to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic retinopathy or | | | |
| diabetic maculopathy prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic nephropathy prior to | , , | , , | , , |
| index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic neuropathy prior to | , , | | . , |
| index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |


| | Empagliflozin | DPP-4 inhibitors | [Country] Study |
|---|---|---|---|
| | at index date | at index date | population |
| | N | N | (Total) |
| History of Diabetic lower limb severe | | | |
| complications prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N(x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of peripheral vascular disease | | | |
| prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N(x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of kidney or genitourinary | | | |
| stones prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of UTI or pyelonephritis prior to | | | |
| index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of liver disease prior to index | | | |
| date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N(x.xx%) |

History of pancreatitis prior to index date

| | Empagliflozin at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of congestive heart failure prior | | | |
| to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of hypertension prior to index | | | |
| date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of stroke prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of myocardial infarction prior to | | | |
| index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of autoimmune disease prior to | | | |
| index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of COPD prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| | | | • • |


| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study population |
|---|---|---|---|
| | N | N | (Total) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Any ICU admission prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Antihypertensives/ diuretics use prior to | | | |
| index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N(x.xx%) | N (x.xx%) | N (x.xx%) |
| NSAIDs use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N(x.xx%) | N (x.xx%) | N (x.xx%) |
| Oral steroids use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Statins/fibrates use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Lipid modifying agents use prior to index | | | |
| date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |


| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Zoledronic acid use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Antibiotic use prior to index date | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| BMI (closest value prior to index date) | | | |
| <20 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 20-24.9 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 25-29.9 | N(x.xx%) | N(x.xx%) | N(x.xx%) |
| >30 | N(x.xx%) | N(x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Smoking status (closest value prior to | | | |
| index date) | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N(x.xx%) | N (x.xx%) | N (x.xx%) |

Alcohol use (closest value prior to index date)


| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| HbA1c in mmol/mol(closest value prior to index date) | | | |
| < 48 (6.5%) mmol/mol | N (x.xx%) | N(x.xx%) | N (x.xx%) |
| ≥ 48 (6.5 %) - <64 mol/mol (8 %) | N (x.xx%) | N(x.xx%) | N (x.xx%) |
| ≥ 64 mmol/mol (8 %) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| eGFR in (mL/min/1.73 m2) | | | |
| <15 (ml/min/1.73 m2) (kidney failure) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 15-29 (ml/min/1.73 m2) (severely decreased) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 30-44 (ml/min/1.73 m2) (Moderately to severely decreased) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 45-59 (ml/min/1.73 m2) (Mildly to moderately decreased) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 60-89 (ml/min/1.73 m2) (Mildly decreased) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥90 (ml/min/1.73 m2) (Normal) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| , , , | ` , | , | • |


| | Empagliflozin<br>at index date | DPP-4 inhibitors<br>at index date | [Country] Study<br>population |
|---|---|---|---|
| | N | N | (Total) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Renal impairment | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Systolic blood pressure | | | |
| < 120 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥120-<139 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥140-<159 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥160 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Diastolic blood pressure | | | |
| < 80 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 80-89 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 90-99 | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 100 or higher | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |

## Boehringer Ingelheim

SEAP for non-interventional study BI Study No: 1245.97


| | Empagliflozin<br>at index date | - 0 | |
|---|---|---|---|
| | N | N | (Total) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |


Table 18 Covariate balance assessment [before/after] matching comparing empagliflozin group to DPP-4 inhibitors group – [Study country].

| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| Age at index (years) | | | | |
| 18-49 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 50-64 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 65-69 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 70-74 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 75-79 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 80-84 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 85 and over | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | <del>-</del> | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| Sex | | | | |
| Male | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Female | N (x.xx%) | N (x.xx%) | | |
| Highest level of education | | | | |
| Compulsory | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Upper secondary | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Post secondary | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Disposable income, individual | | | | |
| < Q1 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| Q1 – Q2 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Q2 - Q3 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| $\geq Q3$ | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| Disposable income, family | NI (v. svat04) | NI (v. vor0/s) | v2 teet p value | std diff |
| < Q1 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Q1 – Q2 | N (x.xx%)<br>N (x.xx%) | N (x.xx%)<br>N (x.xx%) | χ2 test p-value | std diff |
| Q2 – Q3<br>≥ Q3 | N (x.xx%) | N (x.xx%) | χ2 test p-value<br>χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | χ2 test p-varue | sta am |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | 1 | |
| Marital status | | | | |
| Registered partnership (incl. married) | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Widowed | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Separated | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Single | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Calendar year of index date | | | | |
| 2014 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| 2015 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2016 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2017 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2018 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2019 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2020 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2021 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Duration of look-back period | | | - | |
| 1 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 2-5 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 5-9 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 10 and over | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | _ | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | - | |
| Time since first diabetes diagnosis at index da | ate | | | |
| <q1< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>χ2 test p-value</td><td>std diff</td></q1<> | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| ≥Q1- <q2< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>χ2 test p-value</td><td>std diff</td></q2<> | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| ≥Q2- <q3< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>χ2 test p-value</td><td>std diff</td></q3<> | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| ≥Q4 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | - | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| Duration of treated diabetes at index date | | | | |
| Range (min,max) | (min, max) | (min, max) | | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| Diabetes treatment complexity at index date | | | | |
| Monotherapy | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| Dual combination therapy | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Triple combination therapy | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| Insulin use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| Metformin use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| Oral glucose lowering drugs use at index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| Sulfonylureas use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | _ | |

Thiazolidinediones use at index date


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| GLP-1 use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of diabetic complications prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of diabetic retinopathy or diabetic maculopathy prior to index date | | | | |
| Yes | N(x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of diabetic nephropathy prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of diabetic neuropathy prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| History of Diabetic lower limb severe | | | | |
| complications prior to index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of peripheral vascular disease prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of kidney or genitourinary stones prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of UTI or pyelonephritis prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of liver disease prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | _ | |
| History of pancreatitis prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | - | |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| History of congestive heart failure prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N(x.xx%) | | |
| History of hypertension prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of stroke prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of myocardial infarction prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N(x.xx%) | | |
| History of autoimmune disease prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| History of COPD prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |

Any ICU admission prior to index date


| | Empagliflozin users at index date [before/after] matching N DPP-4 inhibitors users at index date [before/after] matching N | | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N(x.xx%) | N(x.xx%) | | |
| Antihypertensives/ diuretics use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N(x.xx%) | N (x.xx%) | _ | |
| NSAIDs use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | _ | |
| Oral steroids use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N(x.xx%) | N (x.xx%) | _ | |
| Statins/fibrates use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| Lipid modifying agents use at index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| Zoledronic acid use at index date | | | | |
| Yes | N(x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| Antibiotic use at index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | | |
| BMI (closest value prior to index date) | | | | |
| <20 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| 20-24.9 | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| 25-29.9 | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| >30 | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| Smoking status (closest value prior to index | | | | |
| date) | | | | |
| Yes | N (x.xx%) | N(x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N(x.xx%) | _ | |
| Alcohol use (closest value prior to index date) | | | | |
| Yes | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| No | N (x.xx%) | N (x.xx%) | _ | |

## Boehringer Ingelheim

SEAP for non-interventional study BI Study No: 1245.97


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | at index date users at index date after] matching [before/after] matching | | Standardized<br>differences |
|---|---|---|---|---|
| HbA1c mmol/mol (closest value prior to index | | | | |
| date) | | | | |
| < 48 (6.5%) mmol/mol | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| ≥ 48 (6.5 %) - <64 mol/mol (8 %) | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| ≥ 64 mmol/mol (8 %) | N (x.xx%) | N (x.xx%) | χ2 test p-value | std diff |
| Range (min,max) | (min, max) | (min, max) | | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| Number of albuminuria tests at index date | | | | |
| Range (min,max) | (min, max) | (min, max) | | |
| mean (± sd) | mean (± sd) | mean (± sd) | t-test p-value | std diff |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | | |
| eGFR in (mL/min/1.73 m2) | | | | |
| <15 (ml/min/1.73 m2) (kidney failure) | N (x.xx%) | N (x.xx%) | N(x.xx%) | N (x.xx%) |
| 15-29 (ml/min/1.73 m2) (severely decreased) | N (x.xx%) | N (x.xx%) | N(x.xx%) | N (x.xx%) |
| 30-44 (ml/min/1.73 m2) (Moderately to severely decreased) | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 45-59 (ml/min/1.73 m2) (Mildly to moderately decreased) | | | | |
| 60-89 (ml/min/1.73 m2) (Mildly decreased) | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥ ( (ml/min/1.73 m2) (Normal) | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |


| | Empagliflozin<br>users at index date<br>[before/after] matching<br>N | DPP-4 inhibitors<br>users at index date<br>[before/after] matching<br>N | P-Value | Standardized<br>differences |
|---|---|---|---|---|
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Renal impairment | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Systolic blood pressure | | | | |
| < 120 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥120-<139 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥140-<159 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥160 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Diastolic blood pressure | | | | |
| < 80 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 80-89 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 90-99 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 100 or higher | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |

Boehringer Ingelheim SEAP for non-interventional study BI Study No: 1245.97


Figure 3 Propensity score distribution in empagliflozin users at index and DPP-4 inhibitors users before matching – [Study country], [Cohort].



Figure 4 Standardized differences for baseline covariates comparing patients using empagliflozin at index and DPP-4 inhibitors users at index date before and after matching – [Study country].

Standardized differences for baseline covariates comparing patients using empagliflozin at index date to patients using [drug group] at index date in the unmatched and matched cohorts – [Country] data



Boehringer Ingelheim SEAP for non-interventional study BI Study No: 1245.97


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Figure 5 Propensity score distribution in non-matched empagliflozin users at index date, matched empagliflozin users at index and matched DPP-4 inhibitors users at index – [Study country], [Cohort].

SEAP for non-interventional study BI Study No: 1245.97




## Boehringer Ingelheim

SEAP for non-interventional study BI Study No: 1245.97


Table 19 Propensity score distribution before and after propensity score matching of empagliflozin users and DPP-4 inhibitors users by decile in [country]

| Propensity score | Decile 1 | Decile 2 | Decile 3 | Decile 4 | Decile 5 | Decile 6 | Decile 7 | Decile 8 | Decile 9 |
|---|---|---|---|---|---|---|---|---|---|
| Before matching | | | | | | | | | |
| Empagliflozin users DPP-4 inhibitors users | X.XXX<br>X.XXX | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx |
| After matching | | | | | | | | | |
| Matched empagliflozin users<br>Matched DPP-4 inhibitors users | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx |


Table 20 Number of patients with incidence of cancer within 12 months after index date

| | Empagliflozin users at index date | DPP-4 inhibitors users at index date |
|---|---|---|
| Number of cancers within 12 months after index date. | N (x.xx%) | N (x.xx%) |

Table 21 TNM staging of [Study outcome] at diagnosis during follow-up after exclusion of cancers occurring within 6 months after index date.

| | [Study outcome] cases in empagliflozin users at index date | [Study outcome] cases<br>in DPP-4 inhibitors<br>users at index date |
|---|---|---|
| TNM staging (T) | | |
| T0 | N (x.xx%) | N (x.xx%) |
| T1 | N (x.xx%) | N (x.xx%) |
| T1a | N (x.xx%) | N (x.xx%) |
| T1b | N (x.xx%) | N (x.xx%) |
| T1c | N (x.xx%) | N (x.xx%) |
| T2 | N (x.xx%) | N (x.xx%) |
| T3 | N (x.xx%) | N (x.xx%) |
| T4 | N (x.xx%) | N (x.xx%) |
| TX | N (x.xx%) | N (x.xx%) |
| NA | N (x.xx%) | N (x.xx%) |
| TNM staging (N) | | |
| N0 | N (x.xx%) | N (x.xx%) |
| N1 | N (x.xx%) | N (x.xx%) |
| NX | N (x.xx%) | N (x.xx%) |
| NA | N (x.xx%) | N (x.xx%) |
| TNM staging (M) | | |
| M0 | N (x.xx%) | N (x.xx%) |
| M1 | N (x.xx%) | N (x.xx%) |
| MX | N (x.xx%) | N (x.xx%) |
| NA | N (x.xx%) | N (x.xx%) |

Table 22 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country/pooled] matched cohort(s). The number of patients in each strata and the total number of person years are also presented.

| Variable | N | N | Person | Rate | Lower | Upper<br>95% Cl |
|---|---|---|---|---|---|---|
| and strata | Patients | events | years | Kate | 95% CI | |
| Absolute incidence | | | | | | |
| Total | N | N | N | X.XX | X.XX | X.XX |
| Exposure category (As | | | | | | |
| treated) | | | | | | |
| Empagliflozin | N | N | N | X.XX | x.xx | x.xx |
| DPP-4 inhibitors | N | N | N | X.XX | x.xx | x.xx |
| Age at index (years) | | | | | | |
| 18-49 | N | N | N | X.XX | X.XX | X.XX |
| 50-64 | N | N | N | X.XX | X.XX | X.XX |
| 65-69 | N | N | N | X.XX | X.XX | X.XX |
| 70-74 | N | N | N | X.XX | X.XX | x.xx |
| 75-79 | N | N | N | X.XX | X.XX | x.xx |
| 80-84 | N | N | N | X.XX | X.XX | X.XX |
| 85 and over | N | N | N | X.XX | X.XX | x.xx |
| Sex | | | | | | |
| Male | N | N | N | X.XX | X.XX | x.xx |
| Female | N | N | N | X.XX | X.XX | x.xx |
| Highest level of education | | | | | | |
| Compulsory | N | N | N | X.XX | X.XX | x.xx |
| Upper secondary | N | N | N | X.XX | X.XX | x.xx |
| Post secondary | N | N | N | X.XX | X.XX | x.xx |
| Disposable income, | · | · | · | | · | · |
| individual | | | | | | |
| < Q1 | N | N | N | X.XX | X.XX | x.xx |
| Q1 – Q2 | N | N | N | X.XX | X.XX | X.XX |
| Q2 – Q3 | N | N | N | X.XX | X.XX | x.xx |
| ≥ Q3 | N | N | N | X.XX | X.XX | X.XX |
| Disposable income, family | - , | - ' | - ' | | | |
| < Q1 | N | N | N | x.xx | X.XX | x.xx |
| Q1 – Q2 | N | N | N | X.XX | X.XX | X.XX |
| Q2 – Q3 | N | N | N | X.XX | X.XX | X.XX |
| ≥ Q3 | N | N | N | X.XX | X.XX | X.XX |


| Variable | N | N | Person | Rate | Lower | Upper |
|---|---|---|---|---|---|---|
| and strata | Patients | events | years | | 95% CI | 95% C |
| Marital status | | | | | | |
| Registered partnership (incl. married) | N | N | N | x.xx | X.XX | x.xx |
| Widowed | N | N | N | X.XX | x.xx | X.XX |
| Separated | N | N | N | X.XX | x.xx | X.XX |
| Single | N | N | N | X.XX | x.xx | x.xx |
| Calendar year of index date | | | | | | |
| 2014 | N | N | N | X.XX | x.xx | X.XX |
| 2015 | N | N | N | X.XX | X.XX | x.xx |
| 2016 | N | N | N | X.XX | X.XX | x.xx |
| 2017 | N | N | N | X.XX | X.XX | x.xx |
| 2018 | N | N | N | X.XX | X.XX | x.xx |
| 2019 | N | N | N | X.XX | x.xx | X.XX |
| 2020 | N | N | N | X.XX | X.XX | X.XX |
| Diabetes treatment<br>complexity at index date | | | | | | |
| | NT | <b>N</b> T | NT | | | |
| Monotherapy | N | N | N | X.XX | X.XX | X.XX |
| Dual combination therapy | N | N | N | X.XX | X.XX | X.XX |
| Triple combination therapy Insulin use | N | N | N | X.XX | X.XX | X.XX |
| Yes | N | N | N | V VV | VVV | v vv |
| No | N | N | N | X.XX | X.XX | X.XX |
| Metformin use | 11 | 11 | 11 | X.XX | X.XX | X.XX |
| Yes | N | N | N | x.xx | x.xx | x.xx |
| No | N | N | N | X.XX | X.XX | x.xx |
| Oral glucose lowering drugs | | - ' | | | | |
| use | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | x.xx |
| Sulfonylureas use | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | x.xx | X.XX |
| Thiazolidinediones use | | | | | | |
| Yes | N | N | N | x.xx | x.xx | x.xx |

| Variable | N | N | Person | Rate | Lower | Upper |
|---|---|---|---|---|---|---|
| and strata | Patients | events | years | Race | 95% CI | 95% C |
| No | N | N | N | X.XX | X.XX | X.XX |
| GLP-1 use | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X,XX | X.XX |
| Diabetic complications | | | | | | |
| Yes | N | N | N | X.XX | x.xx | x.xx |
| No | N | N | N | x.xx | X.XX | x.xx |
| Diabetic retinopathy or diabetic maculopathy | | | | | | |
| Yes | N | N | N | X.XX | x.xx | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Diabetic nephropathy | • | • | · | | | |
| Yes | N | N | N | X.XX | x.xx | X.XX |
| No | N | N | N | X.XX | X,XX | X.XX |
| Diabetic neuropathy | | - ' | - ' | | | |
| Yes | N | N | N | X.XX | X,XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Diabetic lower limb severe | , | - ' | - ' | | | |
| complications | | | | | | |
| Yes | N | N | N | X.XX | X,XX | x.xx |
| No | N | N | N | X.XX | X.XX | x.xx |
| Peripheral vascular disease | | | | | | |
| Yes | N | N | N | x.xx | X.XX | x.xx |
| No | N | N | N | X.XX | X.XX | x.xx |
| Kidney or genitourinary stones | <u> </u> | <u> </u> | <u> </u> | <u> </u> | <u> </u> | · |
| Yes | N | N | N | x.xx | x.xx | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| UTI or pyelonephritis | | | | | | |
| Yes | N | N | N | x.xx | X,XX | x.xx |
| No | N | N | N | X.XX | X.XX | X.XX |
| Liver disease | | | | | | |
| Yes | N | N | N | X.XX | X.XX | x.xx |
| No | N | N | N | X.XX | X.XX | x.xx |

| | Variable<br>and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI |
|---|---|---|---|---|---|---|---|
| Yes | | N | N | N | X.XX | X.XX | X.XX |
| No | | N | N | N | X.XX | X.XX | X.XX |

| Congestive heart failure | | | | | | |
|------------------------------|---|---|---|------|------|------|
| Yes | N | N | N | X,XX | x.xx | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Hypertension | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Stroke | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X,XX |
| Myocardial infarction | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Autoimmune disease | | | | | | |
| Yes | N | N | N | X.XX | x.xx | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| COPD | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Any ICU admission prior to | | | | | | |
| index date | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Antihypertensives/ diuretics | | | | | | |
| use | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X,XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| NSAIDs use | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X,XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Oral steroids | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |

| Variable - | N | N | Person | Rate | Lower | Upper |
|---|---|---|---|---|---|---|
| and strata | Patients | events | years | | 95% CI | 95% CI |
| Statins/fibrates use | | | | | | |
| Yes | N | N | N | X.XX | X,XX | X.XX |
| No | N | N | N | X.XX | X,XX | X.XX |
| Lipid modifying agents use | | | | | | |
| Yes | N | N | N | x.xx | x.xx | x.xx |
| No | N | N | N | X.XX | X.XX | X.XX |
| Zoledronic acid use | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Antibiotic use | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| BMI (closest value prior to index date) | | | | | | |
| <20 | N | N | N | X.XX | X,XX | X.XX |
| 20-24.9 | N | N | N | X.XX | X,XX | X.XX |
| 25-29.9 | N | N | N | x.xx | X.XX | X.XX |
| >30 | N | N | N | X.XX | X.XX | X.XX |
| Smoking status (closest value prior to index date) | | | | | | |
| Yes | N | N | N | X.XX | X,XX | x.xx |
| No | N | N | N | X.XX | X.XX | X.XX |
| Alcohol use (closest value prior to index date) | | | | | | |
| Yes | N | N | N | X.XX | X,XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| HbA1c (closest value prior to index date) | | | | | | |
| < 48 (6.5%) mmol/mol | N | N | N | x.xx | x.xx | x.xx |
| ≥ 48 (6.5 %) - <64 mol/mol (8 %) | N | N | N | X.XX | x.xx | X.XX |
| ≥ 64 mmol/mol (8 %) | N | N | N | X.XX | X.XX | X.XX |
| eGFR in (mL/min/1.73 m2)<br><15 (ml/min/1.73 m2) (kidney<br>failure) | N | N | N | x.xx | x.xx | x.xx |


| Variable | ${f N}$ | N | Person | Rate | Lower | Upper |
|---|---|---|---|---|---|---|
| and strata | Patients | events | years | Rate | 95% CI | 95% CI |
| 15-29 (ml/min/1.73 m2) | N | N | N | 37. 3737 | 37. 3737 | 37 3737 |
| (severely decreased) | IN | 11 | 11 | X.XX | X.XX | X.XX |
| 30-44 (ml/min/1.73 m2) | | | | | | |
| (Moderately to severely | N | N | N | X.XX | X.XX | X.XX |
| decreased) | | | | | | |
| 45-59 (ml/min/1.73 m2) | | | | | | |
| (Mildly to moderately | N | N | N | X.XX | X.XX | X.XX |
| decreased) | | | | | | |
| 60-89 (ml/min/1.73 m2) | NI | NT | Nī | | | |
| (Mildly decreased) | N | N | N | X.XX | X.XX | X.XX |
| ≥90 (ml/min/1.73 m2) | NI | NT | NI | | | |
| (Normal) | N | N | N | X.XX | X.XX | X.XX |
| Renal impairment | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX |
| Systolic blood pressure | | | | | | |
| < 120 | N | N | N | X.XX | X.XX | X.XX |
| ≥120-<139 | N | N | N | X.XX | X.XX | X.XX |
| ≥140-<159 | N | N | N | X.XX | X.XX | X.XX |
| ≥160 | N | N | N | X.XX | X.XX | X.XX |
| Diastolic blood pressure | | | | | | |
| < 80 | N | N | N | X.XX | X.XX | x.xx |
| 80-89 | N | N | N | X.XX | X.XX | x.xx |
| 90-99 | N | N | N | X.XX | X,XX | X.XX |
| 100 or higher | N | N | N | X.XX | x.xx | X.XX |

Figure 6 Kaplan-Meier survival probability estimates for [Outcome name] in the [Study country] matched cohort stratified by exposure using the as treated definition.



Page 129 of

185

Table 23 Crude hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the crude model with the corresponding 95% CI and p-value—As treated

| Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
|---|---|---|---|
| reference | reference | reference | reference |
| x.xxx | x.xxx | X.XXX | X.XXX |
| | ratio<br>reference | ratio 95% CI reference reference | ratio 95% CI 95% CI reference reference reference |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 24 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the base model with the corresponding 95% CI and p-value—As treated exposure definition.

| Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
|---|---|---|---|
| reference | reference | reference | reference |
| X.XXX | X.XXX | X.XXX | x.xxx |
| | ratio<br>reference | ratio 95% CI reference reference | ratio 95% CI 95% CI reference reference reference |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 25 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—As treated exposure definition. [Stratifying variable if any]

| Variables | Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
|---|---|---|---|---|
| AT exposure | | | | |
| DPP-4 inhibitors | reference | reference | reference | reference |
| Empagliflozin | X.XXX | x.xxx | x.xxx | x.xxx |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 26 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—Cumulative dose of empagliflozin exposure definition.

| Variables | Hazard | Lower | Upper | P-value |
|---|---|---|---|---|
| v ariables | ratio | 95% CI | 95% CI | r-varue |
| Cumulative dose of empagliflozin | | | | |
| Never exposed | reference | reference | reference | reference |
| < Q1 | X.XXX | X.XXX | X.XXX | X.XXX |
| Q1 – Q2 | X.XXX | X.XXX | X.XXX | X.XXX |
| Q2 – Q3 | X.XXX | X.XXX | X.XXX | X.XXX |
| ≥ Q3 | X.XXX | X.XXX | X.XXX | X.XXX |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 27 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—daily dose of empagliflozin exposure definition.

| Variables | Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
|---|---|---|---|---|
| Daily dose of empagliflozin | | | | |
| Never exposed | reference | reference | reference | reference |
| 10 mg | X,XXX | X.XXX | X.XXX | x.xxx |
| 25 mg | X.XXX | X.XXX | X.XXX | X.XXX |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 28 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—Cumulative exposure duration to empagliflozin.

| Variables | Hazard | Lower | Upper | P-value |
|---|---|---|---|---|
| | ratio | 95% CI | 95% CI | |
| Cumulative duration of empagliflozin | | | | |
| Never exposed | reference | reference | reference | reference |
| < Q1 | X.XXX | X.XXX | X.XXX | X.XXX |
| Q1 – Q2 | X.XXX | x.xxx | x.xxx | X.XXX |
| Q2 - Q3 | X.XXX | x.xxx | x.xxx | X.XXX |
| ≥ Q3 | X.XXX | X.XXX | X.XXX | X.XXX |

185

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 29 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented.

| Variable and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI |
|---|---|---|---|---|---|---|
| AT exposure | | | | | | |
| DPP-4 inhibitors | N | N | N | X.XX | x.xx | X,XX |
| Empagliflozin | N | N | N | X.XX | x.xx | x.xx |

185

Table 30 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented.

| Variable and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI |
|---|---|---|---|---|---|---|
| Cumulative dose of empagliflozin | | | | | | |
| Never exposed | N | N | N | X.XX | X.XX | X.XX |
| < Q1 | N | N | N | X.XX | X.XX | X.XX |
| Q1 – Q2 | N | N | N | X.XX | X.XX | X.XX |
| Q2 - Q3 | N | N | N | X.XX | X.XX | X.XX |
| $\geq Q3$ | N | N | N | X.XX | X.XX | X.XX |


Table 31 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented.

| Variable | N | N | Person | Rate | Lower | Upper |
|---------------|-----------------|--------|--------|------|--------|--------|
| and strata | <b>Patients</b> | events | years | | 95% CI | 95% CI |
| Daily dose of | | | | | | |
| empagliflozin | | | | | | |
| Never exposed | N | N | N | X.XX | X.XX | X.XX |
| 10mg | N | N | N | X.XX | X.XX | X.XX |
| 25mg | N | N | N | X.XX | x.xx | X.XX |


Table 32 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the [Study country] matched cohort. The number of patients in each strata and the total number of person years are also presented.

| Variable<br>and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI |
|---|---|---|---|---|---|---|
| Cumulative exposure | | | | | | |
| duration to | | | | | | |
| empagliflozin | | | | | | |
| Never exposed | N | N | N | X.XX | X.XX | X.XX |
| < Q1 | N | N | N | X.XX | X.XX | X.XX |
| Q1 – Q2 | N | N | N | X.XX | X.XX | X.XX |
| Q2 - Q3 | N | N | N | X.XX | X.XX | X.XX |
| $\geq Q3$ | | | | | | |
Figure 7. Distribution of the stabilized weights on log scale by time from index date for [drug group]

### Stabilized weights




Table 36. Number of yearly albuminaria tests stratified by exposure group - [Study country]

| | Empagliflozin | DPP-4 inhibitors |
|-----------------|----------------|------------------|
| No. of tests | | |
| 0 | N (x.xx%) | N (x.xx%) |
| 1 | N (x.xx%) | N (x.xx%) |
| 2 | N (x.xx%) | N (x.xx%) |
| More than 2 | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |

Table 37 Patients baseline characteristics in each of the study groups in the UK, stratified by CPRD database.

| | GC | OLD | Au | Aurum |
|---|---|---|---|---|
| | Empagliflozin<br>N = | DPP-4 inhibitors<br>N = | Empagliflozin<br>N = | DPP-4 inhibitors<br>N = |
| Age at index | | | | |
| (years) | | | | |
| 18-49 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 50-64 | N(x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 65-69 | N(x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 70-74 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 75-79 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 80-84 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 85 and over | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Sex | | | | |
| Male | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Female | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Highest level of education Compulsory Upper secondary | N (x.xx%)<br>N (x.xx%) | N (x.xx%)<br>N (x.xx%) | N (x.xx%)<br>N (x.xx%) | N (x.xx%)<br>N (x.xx%) |
| Post secondary | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Disposable income, Individual | , | | | |
| < Q1 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q1 – Q2 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q2 - Q3 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq Q3$ | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Disposable | | | | |
| income, family | | | | |
| < Q1 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q1 – Q2 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Q2 – Q3 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq Q3$ | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |

| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
|---|---|---|---|---|
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Marital status | | | | |
| Registered | | | | |
| partnership (incl. | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| married) | / | / | / | / |
| Widowed | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Separated | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Single | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Calendar year of | | | | |
| index date | <b>N</b> I ( 0() | <b>3.</b> I ( 0() | <b>N</b> I ( 0() | NI ( 0() |
| 2014 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2015 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2016 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2017 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2018 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2019 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2020 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2021 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Duration of look- | | | | |
| back period<br>1 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 2-5 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 6-9 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 10 and over | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | $(\min, \max)$ | (min, max) | $(\min, \max)$ | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3 |
| Time since first | medium (Q1,Q5) | medium (Q1,Q0) | medium (Q1,Q0) | medium (Q1,Q0 |
| diabetes diagnosis | | | | |
| at index date | | | | |
| <q1< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td></q1<> | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq$ (x <q2< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td></q2<> | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| $\geq$ (x <q3< td=""><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td><td>N (x.xx%)</td></q3<> | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| _ (<br>≥( | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean $(\pm sd)$ | , | · | , | |
| | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3 |

| | ger | ingemenn mærnational Ginor | 01 0110 01 111010 01 110 41111140 | - u - c p c |
|---|---|---|---|---|
| Duration of treated diabetes at | | | | |
| index date | | | | |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Diabetes treatment | median (Q1,Q5) | median (Q1,Q5) | illediaii (Q1,Q3) | illediaii (Q1,Q3) |
| complexity at | | | | |
| index date | | | | |
| Monotherapy | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Dual combination | , | , , | , | |
| therapy | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Triple | | | | |
| combination | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| therapy | , | , | , | , |
| Insulin use prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Insulin use at | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Metformin use | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Metformin use at | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Oral glucose | | | | |
| lowering drugs use | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Oral glucose | | | | |
| lowering drugs use | | | | |
| at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |

| roprietary confidential informa | ation © 2024 Roehringer | Ingelheim International GmbF | I or one or more of its affiliat | ed companies |
|---|---|---|---|---|
| Sulfonylureas use | mon © 2024 Documer | mgemenn mæmanonar Gillor | i of one of more of its airillat | ca companies |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Sulfonylureas use | . ( | . ( , | . ( | . ( |
| at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Thiazolidinediones | , | , | , | , |
| use prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Thiazolidinediones | • | • | • | . , |
| use at index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| GLP-1 use prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| GLP-1 use at index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic | | | | |
| complications | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic | | | | |
| retinopathy or | | | | |
| diabetic | | | | |
| maculopathy prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic | | | | |
| nephropathy prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |

| 1 3 | Č | C | | 1 |
|---------------------|-----------|-----------|-----------|-----------|
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of diabetic | | | | |
| neuropathy prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of Diabetic | | | | |
| lower limb severe | | | | |
| complications | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of | | | | |
| peripheral vascular | | | | |
| disease prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of kidney | | | | |
| or genitourinary | | | | |
| stones prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of UTI or | | | | |
| pyelonephritis | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of liver | | | | |
| disease prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of | | | | |
| pancreatitis prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| | | • | • | • |

| Proprietary confidential informa | ation © 2024 Boehringer | Ingelheim International GmbH | I or one or more of its affiliat | ed companies |
|---|---|---|---|---|
| History of | | | | |
| congestive heart | | | | |
| failure prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of | | | | |
| hypertension prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of stroke | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of | | | | |
| myocardial | | | | |
| infarction prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of | | | | |
| autoimmune | | | | |
| disease prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N(x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| History of COPD | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N(x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Any ICU | | | | |
| admission prior to | | | | |
| index date | <b>N</b> T ( 20) | <b>3.</b> 1 ( 2 ( ) | <b>N</b> I ( 2() | NT ( 20) |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |

Antihypertensives/ diuretics use prior to index date


| Proprietary confidential infor | mation © 2024 Boehringer | Ingelheim International GmbH | or one or more of its affiliate | ed companies |
|---|---|---|---|---|
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| NSAIDs use prior | | | | |
| to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Oral steroids use | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Statins/fibrates use | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Lipid modifying | | | | |
| agents use prior to | | | | |
| index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Zoledronic acid | | | | |
| use prior to index | | | | |
| date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Antibiotic use | | | | |
| prior to index date | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| BMI (closest value | | | | |
| prior to index | | | | |
| date) | | | | |
| <20 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 20-24.9 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 25-29.9 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| >30 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q) |

Smoking status (closest value prior to index date)

| | | | 105 | |
|---|---|---|---|---|
| roprietary confidential infor | mation © 2024 Boehringer | Ingelheim International GmbH | or one or more of its affiliat | ed companies |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Alcohol use | | | | |
| (closest value prior | | | | |
| to index date) | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| HbA1c in | | | , , | , , |
| mmol/mol(closest | | | | |
| value prior to | | | | |
| index date) | | | | |
| < 48 (6.5%) | <b>N</b> I ( 0() | <b>3.</b> I ( 0() | <b>N</b> I ( 0() | <b>N</b> T ( 0() |
| mmol/mol | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥ 48 (6.5 %) - <64 | <b>N</b> T ( 0() | <b>3.</b> I ( 0() | <b>N</b> I ( 0() | <b>N</b> I ( 0() |
| mol/mol (8 %) | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥ 64 mmol/mol (8 | <b>N</b> T ( 0() | 3.1 ( 0() | <b>N</b> T ( 2() | <b>N</b> T ( 0() |
| %) | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q |
| eGFR in | ( ( , ( ) | ( ( , ( ) | ( ( ) ( ) | <u> </u> |
| (mL/min/1.73 m2) | | | | |
| <15 (ml/min/1.73 | | | | |
| m2) (kidney | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| failure) | - ( ( / ) | - ' () | - ( ( ) | - · () |
| 15-29 | | | | |
| (ml/min/1.73 m2) | | | | |
| (severely | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| decreased) | | | | |
| 30-44 | | | | |
| (ml/min/1.73 m2) | | | | |
| (Moderately to | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| severely | 1 (A.A. 70) | 1 (A.A.A. / 0) | 11 (A.M. 70) | 11 (A.AA70) |
| decreased) | | | | |
| 45-59 | | | | |
| (ml/min/1.73 m2) | | | | |
| (Mildly to | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| moderately | 1 (M.M. /0) | 1 (A.AA /0) | 1 (A.AA/0) | 11 (A.AA /0) |
| decreased) | | | | |
| 60-89 | | | | |
| | N (x xx%) | N (v vv%) | N (x xx%) | N (x vv%) |
| (Mildly decreased) | 11 (A.AA/0) | 11 (A.AA/U) | 11 (A.AA/U) | 11 (1.11/0) |
| (ml/min/1.73 m2) | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |

| Proprietary confidential infor | mation © 2024 Boehringer I | ngelheim International GmbH | I or one or more of its affiliate | ed companies |
|---|---|---|---|---|
| $\geq$ 90 (ml/min/1.73 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (27 2220/4) |
| m2) (Normal) | IN (X.XX%0) | IN (X.XX%) | IN (X.XX%0) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Renal impairment | | | | |
| Yes | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| No | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Systolic blood | | | | |
| pressure | | | | |
| < 120 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N(x.xx%) |
| ≥120-<139 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥140-<159 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| ≥160 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |
| Diastolic blood | | | | |
| pressure | | | | |
| < 80 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 80-89 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 90-99 | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| 100 or higher | N (x.xx%) | N (x.xx%) | N (x.xx%) | N (x.xx%) |
| Range (min,max) | (min, max) | (min, max) | (min, max) | (min, max) |
| mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) | mean (± sd) |
| median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) | median (Q1,Q3) |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 38 Incidence rates per 1000 patient years of [Outcome name] with 95% confidence interval in the UK-CPRD population stratified by CPRD databases (GOLD and Aurum). The number of patients in each strata and the total number of person years are also presented.

| Variable | GOLD | | | | | | Aurum | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI |
| Absolute | | | | | | | | | | | | |
| incidence | | | | | | | | | | | | |
| Total | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Exposure category | | | | | | | | | | | | |
| (As treated) | | | | | | | | | | | | |
| Empagliflozin | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| DPP-4 inhibitors | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Age at index | | | | | | | | | | | | |
| (years) | | | | | | | | | | | | |
| 18-49 | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 50-64 | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 65-69 | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 70-74 | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 75-79 | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 80-84 | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 85 and over | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Sex | | | | | | | | | | | | |
| Male | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Female | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |


| Variable | GOLD | | | | | Aurum | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI |
| Highest level of | | | • | | | | | | • | | | |
| education | | | | | | | | | | | | |
| Compulsory | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Upper secondary | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Post secondary | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Disposable | | | | | | | | | | | | |
| income, individual | | | | | | | | | | | | |
| < Q1 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Q1 – Q2 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Q2 - Q3 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| ≥ Q3 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Disposable | | | | | | | | | | | | |
| income, family | | | | | | | | | | | | |
| < Q1 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Q1 – Q2 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Q2 - Q3 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| ≥ Q3 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Marital status | | | | | | | | | | | | |
| Registered | | | | | | | | | | | | |
| partnership (incl. married) | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Widowed | N | N | N | x.xx | X.XX | x.xx | N | N | N | X.XX | X.XX | X.XX |


| Variable | | | GOI | ĹD | | | CI Patients events years Rate 95% CI 95% x N N N x.xx x.xx x.xx x N N N < | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI | | | | Rate | | Upper<br>95% CI |
| Separated | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Single | N | N | N | x.xx | X.XX | X,XX | N | N | N | x.xx | X.XX | X.XX |
| Calendar year of | | | | | | | | | | | | |
| index date | | | | | | | | | | | | |
| 2014 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 2015 | N | N | N | x.xx | X.XX | X,XX | N | N | N | x.xx | X.XX | X.XX |
| 2016 | N | N | N | x.xx | X.XX | X,XX | N | N | N | x.xx | X.XX | X.XX |
| 2017 | N | N | N | x.xx | X.XX | X,XX | N | N | N | x.xx | X.XX | X.XX |
| 2018 | N | N | N | x.xx | X.XX | X,XX | N | N | N | x.xx | X.XX | X.XX |
| 2019 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 2020 | N | N | N | x.xx | X.XX | X,XX | N | N | N | x.xx | X.XX | X.XX |
| 2021 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Diabetes treatment complexity at index date | | | | | | | | | | | | |
| Monotherapy | N | N | N | X.XX | X.XX | X,XX | N | N | N | X.XX | X.XX | X.XX |
| Dual combination therapy | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Triple combination therapy | N | N | N | x.xx | X.XX | x.xx | N | N | N | X.XX | X.XX | X.XX |

Insulin use


| Variable | | | GOI | LD | | | % CI Patients events years Nate 95% CI 95% CI X.XX N N N X.XX X.XX X.XX X.XX N N N X.XX X.XX X.XX X.XX N N N X.XX X.XX X.XX X.XX N N N X.XX X.XX X.XX X.XX N N N X.XX X.XX X.XX | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N | N | Person | ъ. | Lower | Upper | N | N | Person | ъ. | Lower | Upper |
| | <b>Patients</b> | events | years | Rate | 95% CI | 95% CI | <b>Patients</b> | events | years | Kate | 95% CI | 95% CI |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Metformin use | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Oral glucose | | | | | | | | | | | | |
| lowering drugs use | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Sulfonylureas use | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Thiazolidinediones | | | | | | | | | | | | |
| use | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| GLP-1 use | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Diabetic | | | | | | | | | | | | |
| complications | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | x.xx | X.XX |


| Variable | | | GOI | ĹD | | | % CI Patients events years Rate 95% CI 95% CI x.xx N N N x.xx x.xx x.xx x.xx N N N x.xx x.xx x.xx x.xx N N N x.xx x.xx x.xx x.xx N N N x.xx x.xx x.xx x.xx N N N x.xx x.xx x.xx | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI | | | | Rate | | Upper<br>95% CI |
| No | N | N | N | X.XX | x.xx | x.xx | | | | X.XX | | X.XX |
| Diabetic | | | | | | | | | | | | _ |
| retinopathy or | | | | | | | | | | | | |
| diabetic | | | | | | | | | | | | |
| maculopathy | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Diabetic<br>nephropathy | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Diabetic | | | | | | | | | | | | |
| neuropathy | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | | | | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Diabetic lower | | | | | | | | | | | | |
| limb severe | | | | | | | | | | | | |
| complications | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Variable | | | GOI | ĹD | | | CI Patients events years Rate 95% CI 95% x N N N x.xx x.xx x x N N N x.xx x.xx x x N N N x.xx x.xx x x N N N x.xx x.xx x x N N N x.xx x.xx x x N N N x.xx x.xx x | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI | | | | Rate | | Upper<br>95% CI |
| Peripheral<br>vascular disease | | | • | | | | | | • | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Kidney or<br>genitourinary<br>stones | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| UTI or pyelonephritis | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | x.xx |
| Liver disease | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Pancreatitis | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |

Congestive heart

failure


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Variable | | | GOI | ĹD | | | CI Patients events years Rate 95% CI 95% CI x N N N x.xx x.xx x.xx x N N N x.xx x.xx x.xx | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N | N | Person | D-4- | Lower | Upper | N | N | Person | D-4- | Lower | Upper |
| | <b>Patients</b> | events | years | Rate | 95% CI | 95% CI | <b>Patients</b> | events | years | Kate | 95% CI | 95% CI |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Hypertension | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Stroke | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Myocardial | | | | | | | | | | | | |
| infarction | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Autoimmune | | | | | | | | | | | | |
| disease | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| COPD | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |

Any ICU

admission prior to

index date


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Variable | | | GOI | ĹD | | | % CI Patients events years Rate 95% CI 95% xx N N N xxx x | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N | N | Person | Rate | Lower | Upper | | N | Person | Rate | | Upper |
| | Patients | events | years | Tute | 95% CI | 95% CI | Patients | events | years | ruce | 95% CI | 95% CI |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Antihypertensives/ | | | | | | | | | | | | |
| diuretics use | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| NSAIDs use | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Oral steroids | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Statins/fibrates use | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Lipid modifying | | | | | | | | | | | | |
| agents use | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |

Zoledronic acid

use


| Variable | | | GOI | ĹD | | | % CI Patients events years Rate 95% CI 95% xx N N N x.xx x.xx x.xx xx N N N x.xx x.xx x.xx | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N<br>Patients | N<br>events | Person<br>years | Rate | Lower<br>95% CI | Upper<br>95% CI | | | | Rate | | Upper<br>95% CI |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Antibiotic use | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| BMI (closest value | | | | | | | | | | | | |
| prior to index | | | | | | | | | | | | |
| date) | | | | | | | | | | | | |
| <20 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 20-24.9 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 25-29.9 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| >30 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | x.xx | X.XX |
| Smoking status | | | | | | | | | | | | |
| (closest value prior | | | | | | | | | | | | |
| to index date) | | | | | | | | | | | | |
| Yes | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Alcohol use | | | | | | | | | | | | |
| (closest value prior | | | | | | | | | | | | |
| to index date) | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | x.xx | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |


| Variable | | | GOI | ĹD | | | 6 CI Patients events years Nate 95% CI 95% xx N N N xxx x | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N | N | Person | Rate | Lower | Upper | N | N | Person | Data | Lower | Upper |
| | Patients | events | years | Kate | 95% CI | 95% CI | Patients | events | years | Kate | 95% CI | 95% CI |
| HbA1c (closest | | | | | | | | | | | | |
| value prior to | | | | | | | | | | | | |
| index date) | | | | | | | | | | | | |
| < 48 (6.5%) | N | N | N | X.XX | x.xx | x.xx | N | N | N | X.XX | x.xx | x.xx |
| mmol/mol | | | | | | | | | | | | |
| ≥ 48 (6.5 %) - <64<br>mol/mol (8 %) | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| ≥ 64 mmol/mol (8 %) | N | N | N | x.xx | x.xx | X.XX | N | N | N | X.XX | x.xx | x.xx |
| eGFR in | | | | | | | | | | | | |
| (mL/min/1.73 m2) | | | | | | | | | | | | |
| <15 | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 15-29 | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| 30-44 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 45-59 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 60-89 | N | N | N | X.XX | X.XX | X.XX | N | N | N | x.xx | X.XX | X,XX |
| ≥90 | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| Renal impairment | | | | | | | | | | | | |
| Yes | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |
| No | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | X.XX |

Systolic blood

pressure

### Boehringer Ingelheim

SEAP for non-interventional study BI Study No: 1245.97


| Variable | | | GO1 | LD | | | | | Aur | um | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and strata | N | N | Person | Data | Lower | Upper | N | N | Person | Data | Lower | Upper |
| | <b>Patients</b> | events | years | Rate | 95% CI | 95% CI | <b>Patients</b> | events | years | Rate | 95% CI | 95% CI |
| < 120 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| ≥120-<139 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| ≥140-<159 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| ≥160 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| Diastolic blood | | | | | | | | | | | | |
| pressure | | | | | | | | | | | | |
| < 80 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X,XX | X.XX |
| 80-89 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X,XX | X.XX |
| 90-99 | N | N | N | x.xx | X.XX | X.XX | N | N | N | x.xx | X.XX | X.XX |
| 100 or higher | N | N | N | X.XX | X.XX | X.XX | N | N | N | X.XX | X.XX | x.xx |


Table 39 Crude hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort, stratified by databases. The table shows the hazard ratios (HRs) using the crude model with the corresponding 95% CI and p-value—As treated

| | | GC | OLD | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|
| | Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value | Hazard ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
| AT exposure | | | | | | | | |
| DPP-4 inhibitors | reference | reference | reference | reference | reference | reference | reference | reference |
| Empagliflozin | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 40 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort, stratified by databases. The table shows the hazard ratios (HRs) using the base model with the corresponding 95% CI and p-value—As treated

| | | GC | OLD | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|
| | Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value | Hazard ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
| AT exposure | | | | | | | | |
| DPP-4 inhibitors | reference | reference | reference | reference | reference | reference | reference | reference |
| Empagliflozin | X.XXX | X.XXX | X.XXX | X.XXX | x.xxx | X.XXX | X.XXX | X.XXX |
| inhibitors | | | | | | | | |


Table 41 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort, stratified by databases. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—As treated

| | | GC | OLD | | | Aurum | | |
|---|---|---|---|---|---|---|---|---|
| | Hazard<br>ratio | Lower<br>95% CI | Upper<br>95% CI | P-value | Hazard ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
| AT exposure | | | | | | | | |
| DPP-4 inhibitors | reference | reference | reference | reference | reference | reference | reference | reference |
| Empagliflozin | x.xxx | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |

SEAP for non-interventional study BI Study No: 1245.97


Table 42 Crude hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort after adding CPRD database as a stratification variable. The table shows the hazard ratios (HRs) using the crude model with the corresponding 95% CI and p-value—As treated

| | | Country- UK | | |
|---|---|---|---|---|
| | Hazard ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
| AT exposure | | | | |
| DPP-4 inhibitors | reference | reference | reference | reference |
| Empagliflozin | x.xxx | X.XXX | X.XXX | X,XXX |

SEAP for non-interventional study BI Study No: 1245.97


Table 43 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the UK matched cohort after adding CPRD database as a stratification variable. The table shows the hazard ratios (HRs) using the base model with the corresponding 95% CI and p-value—As treated exposure definition.

| Hazard ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
|---|---|---|---|
| reference | reference | reference | reference |
| X.XXX | X.XXX | X.XXX | x.xxx |
| | reference | reference reference | reference reference reference |

Boehringer Ingelheim

SEAP for non-interventional study BI Study No: 1245.97


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 44 Adjusted hazard ratios for [Outcome Name] incidence estimated using the Cox proportional hazards model in the [Study country] matched cohort after adding CPRD database as a stratification variable. The table shows the hazard ratios (HRs) using the adjusted model with the corresponding 95% CI and p-value—As treated exposure definition.

| Variables | Hazard ratio | Lower<br>95% CI | Upper<br>95% CI | P-value |
|---|---|---|---|---|
| AT exposure DPP-4 inhibitors Empagliflozin | reference | reference | reference | reference |
| | x.xxx | x.xxx | x.xxx | x.xxx |

Figure 8. Meta-analysis of [hazard/odds] ratios of [outcome] for the [analysis type] using a random-effects model

| | N Events (IR/100 | 00 PY) | | | | | Average PY | |
|---|---|---|---|---|---|---|---|---|
| Study E | Empagliflozin | DPP-4 | | Weights | Effect size [95% CI] | N | Empagliflozin | DPP-4 |
| CPRD | N (N) | N (N) | | N % | N [N, N] | N | N | N |
| Sweden | N (N) | N (N) | - | N % | N [N, N] | N | N | N |
| Finland | N (N) | N (N) | | N % | N [N, N] | N | N | N |
| Meta analysis (ra | indom effects) | | 0.71 0.91 1.11 | N % | N [N, N] | N | N | N |
| | | | | .1 | | | | |
| | | | Hazard Ratio (log scale | 5) | | | | |

#### Random effects model:

Heterogeneity: Q (df: N) = N, p-value N, I<sup>2</sup> = N% [N%, N%], τ<sup>2</sup> = N [N, N].

Figure 9. Meta-analysis of hazard ratios of [outcome] for the as-treated analysis of empaglifozin users vs DPP-4 users using a fixed-effect model (sensitivity analysis)

| tudy | | 00 PY) | | | | | Average | PY |
|---|---|---|---|---|---|---|---|---|
| | Empagliflozin | DPP-4 | | Weights | Effect size [95% CI] | N | Empagliflozin | DPP-4 |
| CPRD | N (N) | N (N) | | N % | N [N, N] | N | N | N |
| Sweden | N (N) | N(N) | - | N % | N [N, N] | Ν | N | N |
| Finland | N (N) | N (N) | | N % | N [N, N] | N | N | N |
| Meta analysis (fixed effects) | | | - | N % | N [N, N] | | | N |
| Meta analysis (r | random effects) | | | N % | N [N, N] | N N | | |

#### Fixed effects model:

Overall effect: Z = N, p-value N.

Figure 10. Average number of diabetes-related healthcare visits per patient recorded in the source population for study years 2015-[end of study year]



Figure 11. Number of monthly incident users in [Year] for empaglifozin and DPP-4 inhibitors for [Study country]



Figure 12. Number of quarterly incident users in [year] for empaglifozin and DPP-4 inhibitors for [Study country]



Figure 13. Number of incident users of each study drug group for each study year in [Study country].



Figure 14. Average number (95% CIs) of prescriptions per patient in the source population in [Study country] per quarter from January 2015 to December [End of study year]



185

Table 45. Incidence rate of urinary tract cancer in the source population for all study years from 2015 to end of study year.

| Country and study year | N of patients | N of events | Person<br>years | Incidence<br>rate | Lower<br>95% CI | Upper<br>95% CI |
|---|---|---|---|---|---|---|
| [Study country] | | | | | | |
| 2015 | N | N | N | x.xx | X.XX | X.XX |
| 2016 | N | N | N | X.XX | X.XX | X.XX |
| 2017 | N | N | N | X.XX | X.XX | X.XX |
| 2018 | N | N | N | X.XX | X.XX | X.XX |
| 2019 | N | N | N | X.XX | X.XX | X.XX |
| 2020 | N | N | N | X.XX | X.XX | X.XX |
| 2021 | N | N | N | X.XX | X.XX | X.XX |

## **Annex IV**

# List of drug dosages for empagliflozin, DPP-4 inhibitors and metformin

List of drug dosages extracted from registries in Finland and Sweden:

